CLINICAL TRIAL: NCT01610492
Title: BEL116472. A 2 Year Mechanistic Study of Belimumab in Idiopathic Membranous Glomerulonephropathy
Brief Title: A Study of Belimumab in Idiopathic Membranous Glomerulonephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116472
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Glomerulonephritis, Membranous
Keywords: IMGN; anti-PLA2R antibodies; pharmacokinetics; belimumab; Benlysta; Idiopathic Membranous Glomerulonephropathy; safety; GSK1550188; Lymphostat-B; membrane attack complex
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — belimumab

ARMS (1):
- Cohort 1 (Experimental): 10mg/kg belimumab intravenous (IV) administered at weeks 0 and 2, and then every 4 weeks, over a 24-week treatment period, resulting in a total of 8 doses, and will be assessed for the primary endpoint at week 28. Subjects will then enter the long term phase of the study and receive 10mg/kg belimumab every 4 weeks until week 100,or until they have been in complete remission for at least 3 months, resulting in up to 27 doses.
  Interventions: Drug: belimumab

INTERVENTIONS:
Drug: belimumab — 10mg/kg administered intravenously

SUMMARY:
This is a phase II, open label, experimental medicine study to evaluate the efficacy, safety and mechanism of action of belimumab in subjects with antiphospholipase A2 receptor (PLA2R) autoantibody positive idiopathic membranous glomerulonephropathy (IMGN), and to profile the relationship between biomarkers, autoantibody status and clinical response. 10 milligrams per kilogram (mg/kg) belimumab intravenous (IV) will be administered at weeks 0, 2, and then every 4 weeks, over a 24-week treatment period in subjects with anti-PLA2R antibody positive IMGN followed by a further long term treatment period until subjects reach remission of proteinuria, up to a maximum of 2 years total treatment. All subjects will receive background supportive therapy throughout the study. The dosing frequency will be adjusted to every 2 weeks if the subject's proteinuria as assessed by urinary protein creatinine ratio (PCR) is greater than 1000 milligrams per millimole (mg/mmol) [greater than 10 grams(g)/24 hours (h)], to compensate for loss of belimumab in the urine. Effects on mechanistic markers will be measured by the level of proteinuria, levels of anti-PLA2R antibodies, and various other measures of kidney function. These will be compared to historical data. The pharmacokinetics of belimumab will be measured to confirm dosing in heavily proteinuric subjects. Pharmacodynamic (PD) markers, biomarkers and Quality of Life(QoL) in IMGN subjects will also be investigated. Safety will be assessed by adverse events (AE), clinical laboratory evaluations, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Age & Gender: Male or female between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Histological diagnosis: Have clinical diagnosis of IMGN, as verified by biopsy (either by light microscope with immuno-fluorescence, or by electron microscope) in the last 7 years with non-active disease >3 years (non-active defined as subject not on immunosuppressants and proteinuria <2g per 24h) (biopsy results and slides should be available for independent evaluation).
* Autoantibody: Have positive anti-PLA2R autoantibody test results at screening.
* Proteinuria: Have clinically active disease (nephrotic range proteinuria) for at least 3 months prior to screening and no improvement (less than 30% reduction), despite supportive therapy (which should include maximal tolerated doses of ACE inhibitor or ARB unless contraindicated, and may include statins, diuretics, dietary salt restriction). During screening proteinuria must be greater than 400mg/mmol by PCR (or greater than 4.0g per 24h) as measured from a 24 h urine collection and/or spot urine sample (early morning where possible) on 2 occasions at least 7 days apart.
* Female Subjects: A female subject is eligible to participate if she is not pregnant or nursing and at least one of the following conditions apply: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 Milli-International Units per millilitre(MlU/mL) and estradiol less than 40 picograms per milliliter (less than 147 picomoles per liter) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT.

Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 16 weeks after the last dose

Exclusion Criteria:

* Non-Idiopathic membranous glomerulonephropathy (MGN) or other condition affecting the kidney: If the diagnosis of MGN is secondary to other conditions, or the subject has renal impairment from a condition that is not MGN.
* Severely reduced or deteriorating kidney function: An eGFR at screening < 40 millilitres (mL) /minute (min) /1.73 meter (m)^2 (as determined by 4 variable version Modification of Diet in Renal Disease equation) or kidney function not stable (as defined by > 15% decrease in eGFR in 3 months before screening, unless due to medication change).
* Blood Pressure: Uncontrolled hypertension defined as blood pressure (BP) greater than 150/90 millimeters of mercury (mm Hg) (treatment target greater than and equal to 140/80) as assessed by either : Blood pressures measured 3 times on each of at least 2 clinic visits during screening, after the patient has sat quietly for at least 5 minutes, with greater than 50% of measurements being greater than 150/90 or average daytime blood pressure on a 24 hour ambulatory blood pressure monitor.
* Prior Therapy: Have received treatment with the following therapies at the times specified prior to Day 0: Therapy - B-cell targeted therapy except rituximab (e.g., other anti- CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], B lymphocyte stimulator-receptor fusion protein [BR3], transmembrane activator and calcium modulator and cyclophylin ligand interactor Fc, or belimumab), Time period: anytime; Therapy: Rituximab (Subjects with rituximab treatment between 1 and 2 years prior to Day 0 are eligible if there is documented evidence of B-cell repopulation to >50% of pre-treatment levels.), Period: 2 years; Therapy: Abatacept and any other biologic investigational agent other than B cell targeted therapy (i.e. not approved for sale in the country in which it is being used), Time Period: 364 days; Therapy: Cyclophosphamide or chlorambucil 3 or more courses of systemic corticosteroids for concomitant conditions (e.g., asthma, atopic dermatitis). (Topical or inhaled steroids are permitted.), Time Period: 180 days; Therapy: Anti-tumour necrosis factor (TNF) or anti-IL-6 therapy (e.g. adalimumab, etanercept, infliximab, tocilizumab). Interleukin-1 receptor antagonists (e.g. anakinra). Other immunosuppressive/immunomodulatory agents (e.g azathioprine, 6-mercaptopurine, mycophenolate mofetil (PO)/ mycophenolate mofetil hydrochloride (IV), mycophenolate sodium (PO), methotrexate, tacrolimus, sirolimus, thalidomide, leflunomide, mizoribine, ciclosporin). Intravenous immunoglobulin (IVIG). Plasmapheresis, leukapheresis, Time Period: 90 days; Therapy: A non-biologic investigational agent (i.e. not approved for sale in the country in which it is being used). Intravenous corticosteroid, Adrenocorticotropic hormone (ACTH). Adenocorticotropic hormone (ACTH), aliskiren A change in dose of >50% for angiotensin pathway antihypertensive (e.g., ACE inhibitor, angiotensin receptor blocker), Time Period: 60 days; Therapy: A live vaccine. Greater than 30 milligrams per day (mg/day) corticosteroid, Time Period: 30 days; Therapy: Greater than 10mg/day corticosteroid. A change in dose of a corticosteroid. Note: Changes to inhaled steroids and new topical immunosuppressive agents (e.g., eye drops, topical creams) are allowed, Time Period: 14 days;
* Transplantation: Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Cancer: Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infection: Have required management of acute or chronic infections, as follows: Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria); Hospitalisation for treatment of infection within 60 days prior to Day 0; Use of parenteral (IV or intramuscular) antibiotics (anti-bacterials, anti-virals, anti-fungals, or anti-parasitic agents) within 60 days prior to Day 0.
* Liver disease: Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Other diseases/conditions: Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to IMGN (i.e., cardiovascular, pulmonary, haematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.

or Have a planned surgical procedure or a history of any other medical disease (e.g. cardiopulmonary), laboratory abnormality, or condition (e.g. poor venous access) that, in the opinion of the investigator, makes the subject unsuitable for the study.

* Positive serology: Have a historically positive human immunodeficiency virus (HIV) test or test positive at screening for HIV. Serologic evidence of Hepatitis B (HB) infection based on the results of testing for hepatitis B surface (antigen) (HBsAg), anti-HBc and anti-HBs as follows:- Patients positive for HBsAg are excluded: Patients negative for HBsAg and anti-HBc antibody but positive for anti-HBs antibody and with no history of Hepatitis B vaccination are excluded; Patients negative for HBsAg but positive for both anti-HBc and anti-HBs antibodies are excluded; Patients negative for HBsAg and anti-HBs antibody but positive for anti-HBc antibody are excluded. Positive test for Hepatitis C antibody confirmed on the same sample with a Hepatitis C Recombinant Immunoblot Assay (RIBA) immunoblot assay if available. Subjects who are positive for Hepatitis C antibody and who have a positive or indeterminate result when the Hepatitis C RIBA immunoblot assay is performed on the same sample, or where the Hepatitis C RIBA assay is not available, will not be eligible to participate.
* Liver function tests: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater than and equal to 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin greater than 1.5xULN (isolated bilirubin greater than 1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Immunodeficiency: Have an IgA deficiency [immunoglobulin (Ig)A level < 10 milligrams per deciliter (mg/dL)] or have IgG level < 250 mg/dL and have previously received any non-glucocorticoid immunosuppression during the previous 6 months.
* Laboratory test abnormalities: Have clinically significant abnormalities in screening laboratory assessments (not related to the disease), as judged by investigator.
* Drug sensitivity / Anaphylaxis: History of sensitivity or intolerance to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. History of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Substance abuse: Evidence of current drug or alcohol abuse or dependence.
* Blood donation: Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07-01; Primary Completion 2014-09-24 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United Kingdom (8):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Reading
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Whitechapel, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from July 2012 until March 2014, into this 2 part study of a initial treatment phase, a long term treatment phase, and then followed up for a further 6 months. Results have previously been presented for the initial treatment phase, up to the Week 28 and are now presented for the completed study.
Pre-assignment Details: Screening occurred within 35 days and no less than 14 days before the first scheduled study treatment dose. Total 21 participants were screened; 14 were randomized and entered the initial treatment phase while 11 participants entered the long-term treatment phase. Common reasons for screen failures were insufficient, or improvements in proteinuria.
Groups:
- Belimumab 10 mg/kg IV: Participants received 10 milligrams per kilogram (mg/kg) belimumab intravenous (IV) infusion at Week 0 Week 2 and Week 4, then every 4 weeks over 24 weeks. Participants then entered the long-term phase of the study and received belimumab 10 mg/kg every 4 weeks up to Week 100 or until complete remission had been achieved.
Period: Overall Study
Arm/Group | Belimumab 10 mg/kg IV
Started | 14
Completed | 8
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3
Not completed — Other: Reached stopping criteria | 1
Not completed — Other:Treatment stopped due to remission | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Central/South Asian Heritage | 4
  White- White/Caucasian/European Heritage | 9
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Proteinuria Levels at Week 28
Description: Proteinuria based on urinary protein creatinine ratio (PCR) was measured from 2 consecutive 24 hour (h) urine collection pre and post dosing at Baseline and Week 28 and the mean PCR was determined at each time point. Baseline is defined as the mean of the pre and post dosing Day 0 values. The ratio is defined as the Week 28 value divided by the Baseline value. Ratio to Baseline: Estimated value = 0.76, 2-sided 95% confidence interval (CI)=0.57 to 1.01. The geometric mean method was used to calculate the CI. The analysis was performed on Intent-to-treat (ITT) Population which comprised of all eligible participants who received at least one dose of investigational drug. Only those participants available at the indicated time point (Week 28) were analyzed.
Time Frame: Baseline and Week 28
Population: Intent-to-Treat (ITT) Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 11
Ratio | 0.7552 (45.0)
Statistical Analysis 1: Comparison: Belimumab 10 mg/kg IV; Test type: Other; Geometric Mean = 0.76, 95% CI 2-sided [0.57 to 1.01]

2. Primary Outcome: Change From Baseline in Anti-phospholipase A2 Receptor (PLA2R) Autoantibody Titers at Week 28
Description: PLA2R autoantibody titers in serum were analyzed at Baseline and Week 28 by means of a validated anti- PLA2R enzyme linked immunosorbent assay (ELISA) from EuroImmun. Baseline is defined as the Day 0 value and change from Baseline was calculated as ratio to Baseline by dividing the Week 28 values with the Baseline values. Ratio to Baseline: Estimated value = 0.27, 2-sided 95% CI=0.12 to 0.58. The geometric mean method was used to calculate the CI.
Time Frame: Baseline and Week 28
Population: ITT Population. Only those participants available at the indicated time point (Week 28) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 11
Ratio | 0.2666 (171.0)
Statistical Analysis 1: Comparison: Belimumab 10 mg/kg IV; Test type: Other; Geometric Mean = 0.27, 95% CI 2-sided [0.12 to 0.58]

3. Secondary Outcome: Proteinuria Levels at the Indicated Time Points
Description: Proteinuria based on urinary protein creatinine ratio (PCR) measured from 2 consecutive 24h urine collections at Baseline and Week 28, from a pre-intervention spot urine sample and 24 hour urine collection after visit at Weeks 12, 52, 76 and 104, and from a spot urine sample at week 128. Mean PCR was calculated at each time point where there were 2 samples. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Week 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per millimole (mg/mmol)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
milligrams per millimole (mg/mmol)
  Baseline, n=14 | 724.3157 (40.2)
  Week 12, n=13: number analyzed (Participants) | 13
  Week 12, n=13 | 670.8655 (46.9)
  Week 28, n=11: number analyzed (Participants) | 11
  Week 28, n=11 | 498.1255 (40.9)
  Week 52, n=9: number analyzed (Participants) | 9
  Week 52, n=9 | 356.4209 (174.8)
  Week 76, n=8: number analyzed (Participants) | 8
  Week 76, n=8 | 274.9714 (70.4)
  Week 104, n=10: number analyzed (Participants) | 10
  Week 104, n=10 | 129.9761 (186.0)
  Week 128, n=9: number analyzed (Participants) | 9
  Week 128, n=9 | 75.2359 (136.4)

4. Secondary Outcome: Change From Baseline in Proteinuria Levels at the Indicated Time Points
Description: Proteinuria based on urinary protein creatinine ratio (PCR) measured from 2 consecutive 24h urine collections at Baseline and Week 28, from a pre-intervention spot urine sample and 24 hour urine collection after visit at Weeks 12, 52, 76 and 104, and from a spot urine sample at week 128. Mean PCR was calculated at each time point where there were 2 samples. Baseline is defined as Day 0 value and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Week 12, 28, 52, 76, 104 and Week 128/6 month follow up
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 0.9437 (39.3)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 0.7552 (45.0)
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | 0.5297 (206.7)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 0.4177 (54.3)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 0.1874 (189.3)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 0.1118 (139.1)

5. Secondary Outcome: Anti-phospholipase A2 Receptor (PLA2R) Autoantibody Levels at Indicated Time Points
Description: Anti-PLA2R autoantibody titers in serum were analyzed by means of a validated anti-PLA2R enzyme linked immunosorbent assay (ELISA) assay from Euroimmun. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Week 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: relative units per milliliter (RU/mL)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
relative units per milliliter (RU/mL)
  Baseline, n=14 | 168.3 (138.9)
  Week 12, n=13: number analyzed (Participants) | 13
  Week 12, n=13 | 91.0 (200.4)
  Week 28, n=11: number analyzed (Participants) | 11
  Week 28, n=11 | 46.4 (319.6)
  Week 52, n=9: number analyzed (Participants) | 9
  Week 52, n=9 | 12.9 (358.4)
  Week 76, n=8: number analyzed (Participants) | 8
  Week 76, n=8 | 7.5 (140.4)
  Week 104, n=10: number analyzed (Participants) | 10
  Week 104, n=10 | 3.7 (72.7)
  Week 128, n=8: number analyzed (Participants) | 8
  Week 128, n=8 | 4.4 (112.0)

6. Secondary Outcome: Change From Baseline in Anti-PLA2R Autoantibody Titers at the Indicated Time Points
Description: Anti-PLA2R autoantibody titers in serum were analyzed by means of a validated anti- PLA2R enzyme linked immunosorbent assay (ELISA) from Euroimmun. Baseline is defined as the Day 0 value and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128.
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 0.5362 (58.1)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 0.2666 (171.0)
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | 0.0737 (130.3)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 0.0436 (102.8)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 0.0212 (169.1)
  Week 128; n= 8: number analyzed (Participants) | 8
  Week 128; n= 8 | 0.0284 (243.7)

7. Secondary Outcome: Number of Participants With Complete or Partial Remission
Description: Complete remission is defined as PCR <30 mg/mmol (proteinuria <0.3grams [g]/24 h) with no worsening in renal function (estimated glomerular filtration rate [eGFR] reduction from Baseline <15 percent). Partial remission is defined as PCR <350 mg/mmol (proteinuria <3.5 g/24 h) but >= 30 mg/mmol (proteinuria >= 0.3g/24h) and decrease of >50 percent from Day 0 Baseline, together with no consistent worsening in renal function (eGFR reduction from Baseline <15percent). Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Week 12; Partial remission; n= 13: number analyzed (Participants) | 13
  Week 12; Partial remission; n= 13 | 0
  Week 12; Complete remission; n= 13: number analyzed (Participants) | 13
  Week 12; Complete remission; n= 13 | 0
  Week 28; Partial remission; n= 11: number analyzed (Participants) | 11
  Week 28; Partial remission; n= 11 | 1
  Week 28; Complete remission; n= 11: number analyzed (Participants) | 11
  Week 28; Complete remission; n= 11 | 0
  Week 52; Partial remission; n= 9: number analyzed (Participants) | 9
  Week 52; Partial remission; n= 9 | 2
  Week 52; Complete remission; n= 9: number analyzed (Participants) | 9
  Week 52; Complete remission; n= 9 | 1
  Week 76; Partial remission; n= 8: number analyzed (Participants) | 8
  Week 76; Partial remission; n= 8 | 3
  Week 76; Complete remission; n= 8: number analyzed (Participants) | 8
  Week 76; Complete remission; n= 8 | 0
  Week 104; Partial remission; n= 10: number analyzed (Participants) | 10
  Week 104; Partial remission; n= 10 | 6
  Week 104; Complete remission; n= 10: number analyzed (Participants) | 10
  Week 104; Complete remission; n= 10 | 1
  Week 128; Partial remission; n= 9: number analyzed (Participants) | 9
  Week 128; Partial remission; n= 9 | 6
  Week 128; Complete remission; n= 9: number analyzed (Participants) | 9
  Week 128; Complete remission; n= 9 | 1

8. Secondary Outcome: Time to Complete or Partial Remission
Description: Time to complete or partial remission was estimated using the Kaplan-Meier method. Complete remission is defined as PCR <30 mg/mmol (proteinuria <0.3g/24 h) with no worsening in renal function (eGFR reduction from Baseline <15 percent ). Partial remission is defined as PCR <350 mg/mmol (proteinuria <3.5 g/24 h) but >= 30 mg/mmol (proteinuria >= 0.3g/24h) and decrease of >50 percent from Day 0 Baseline, together with no consistent worsening in renal function (eGFR reduction from Baseline <15 percent). Only 1 participant reached complete remission. Hence, statistical analysis for complete remission was not performed.
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Weeks | 68.20 [28.00 to 93.60]

9. Secondary Outcome: Duration of Complete or Partial Remission
Description: Complete remission is defined as PCR <30 mg/mmol (proteinuria <0.3g/24 h) with no worsening in renal function (eGFR reduction from Baseline <15percent). Partial remission is defined as PCR <350 mg/mmol (proteinuria <3.5 g/24 h) but >= 30 mg/mmol (proteinuria >= 0.3g/24h) and decrease of >50% from Day 0 Baseline, together with no consistent worsening in renal function (eGFR reduction from Baseline <15percent). Only those participants available at the specified time points were analyzed (represented by n=X in category titles). NA indicates that data was not available as only 1 participant reached complete remission. Hence, standard deviation for complete remission was not calculated.
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Days
  Complete remission; n= 1: number analyzed (Participants) | 1
  Complete remission; n= 1 | 365.0 (NA) — NA indicates that data was not available as only 1 participant reached complete remission. Hence, standard deviation for complete remission was not calculated.
  Partial remission; n= 9: number analyzed (Participants) | 9
  Partial remission; n= 9 | 378.6 (186.15)

10. Secondary Outcome: Number of Participants With PLA2R Autoantibody Remission
Description: Incidence of anti-PLA2R autoantibody remission were evaluated by full response and partial response. Full response is defined as antibody undetectable, partial response is defined as reduction in titers by 50 percent. For anti PLA2R autoantibody data, log transformation was applied before the formal analyses. Anti-PLA2R autoantibody blood samples were evaluated at Week 12, 28, 52, 76, 104 and 128/6 week post last-dose. Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Week 12; full response; n= 13: number analyzed (Participants) | 13
  Week 12; full response; n= 13 | 1
  Week 12; partial response; n= 13: number analyzed (Participants) | 13
  Week 12; partial response; n= 13 | 3
  Week 28; full response; n= 11: number analyzed (Participants) | 11
  Week 28; full response; n= 11 | 3
  Week 28; partial response; n= 11: number analyzed (Participants) | 11
  Week 28; partial response; n= 11 | 6
  Week 52; full response; n= 9: number analyzed (Participants) | 9
  Week 52; full response; n= 9 | 4
  Week 52; partial response; n= 9: number analyzed (Participants) | 9
  Week 52; partial response; n= 9 | 5
  Week 76; full response; n= 8: number analyzed (Participants) | 8
  Week 76; full response; n= 8 | 4
  Week 76; partial response; n= 8: number analyzed (Participants) | 8
  Week 76; partial response; n= 8 | 4
  Week 104; full response; n= 10: number analyzed (Participants) | 10
  Week 104; full response; n= 10 | 10
  Week 104; partial response; n= 10: number analyzed (Participants) | 10
  Week 104; partial response; n= 10 | 0
  Week 128; Full response; n= 8: number analyzed (Participants) | 8
  Week 128; Full response; n= 8 | 8
  Week 128; partial response; n= 8: number analyzed (Participants) | 8
  Week 128; partial response; n= 8 | 0

11. Secondary Outcome: Time to Anti-PLA2R Autoantibody Remission
Description: Time to anti-PLA2R autoantibody remission was estimated using Kaplan-Meier method for full response and partial response full response with antibody undetectable and partial response with reduction in titers by 50 percent.
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Weeks
  Partial response | 16.20 [8.00 to 24.00]
  Complete response | 82.00 [16.00 to 92.00]

12. Secondary Outcome: Number of Participants With Anti-PLA2R Autoantibody Relapse
Description: Incidence of anti-PLA2R autoantibody relapse defined as antibody detectable after previously undetectable. Anti-PLA2R autoantibody blood samples were evaluated at Week 12, 28, 52, 76, 104/4 week post last dose, Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 0
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 0
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | 0
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 0
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 0
  Week 128; n= 8: number analyzed (Participants) | 8
  Week 128; n= 8 | 0

13. Secondary Outcome: eGFR Levels at the Indicated Time Points
Description: eGFR was assessed from levels of creatinine using the 4 variable version of the modification of diet in renal disease (MDRD) equation as recommended by National Kidney Foundation-Chronic Kidney Disease (NKF-CKD) guidelines. Baseline for eGFR is defined as the mean of the screening and Day 0 values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up.
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min/1.73meter^2)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
milliliter/minute (mL/min/1.73meter^2)
  Baseline; n= 14 | 69.8170 (32.9)
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 66.2639 (35.4)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 65.0866 (36.1)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 65.1308 (45.0)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 61.6732 (47.1)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 69.7692 (39.1)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 64.7984 (39.2)

14. Secondary Outcome: Change From Baseline in eGFR Levels at the Indicated Time Points
Description: eGFR was assessed from levels of creatinine using the 4 variable version of the modification of diet in renal disease (MDRD) equation as recommended by national kidney foundation-chronic kidney disease (NKF-CKD) guidelines. Baseline for eGFR is defined as the mean of the Screening and Day 0 values and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  Week 2, n=14 | 0.9954 (10.8)
  Week 4, n= 13: number analyzed (Participants) | 13
  Week 4, n= 13 | 0.9190 (16.4)
  Week 8, n= 13: number analyzed (Participants) | 13
  Week 8, n= 13 | 0.9035 (16.2)
  Week 12, n= 13: number analyzed (Participants) | 13
  Week 12, n= 13 | 0.9339 (17.1)
  Week 16, n= 12: number analyzed (Participants) | 12
  Week 16, n= 12 | 0.9521 (12.5)
  Week 20, n= 8: number analyzed (Participants) | 8
  Week 20, n= 8 | 0.9819 (11.8)
  Week 24, n= 11: number analyzed (Participants) | 11
  Week 24, n= 11 | 0.9274 (17.1)
  Week 28, n= 11: number analyzed (Participants) | 11
  Week 28, n= 11 | 0.9694 (21.1)
  Week 32, n= 9: number analyzed (Participants) | 9
  Week 32, n= 9 | 1.0099 (19.5)
  Week 36, n= 11: number analyzed (Participants) | 11
  Week 36, n= 11 | 0.9692 (17.4)
  Week 40, n= 11: number analyzed (Participants) | 11
  Week 40, n= 11 | 0.9425 (20.8)
  Week 44, n= 10: number analyzed (Participants) | 10
  Week 44, n= 10 | 0.9531 (22.6)
  Week 48, n= 8: number analyzed (Participants) | 8
  Week 48, n= 8 | 0.9929 (23.8)
  Week 52, n= 7: number analyzed (Participants) | 7
  Week 52, n= 7 | 0.9290 (27.7)
  Week 56, n= 9: number analyzed (Participants) | 9
  Week 56, n= 9 | 1.0181 (21.9)
  Week 60, n= 9: number analyzed (Participants) | 9
  Week 60, n= 9 | 0.9805 (26.8)
  Week 64, n=9: number analyzed (Participants) | 9
  Week 64, n=9 | 1.0217 (23.5)
  Week 68, n=8: number analyzed (Participants) | 8
  Week 68, n=8 | 1.0233 (24.6)
  Week 72, n=8: number analyzed (Participants) | 8
  Week 72, n=8 | 1.0168 (28.3)
  Week 76, n=8: number analyzed (Participants) | 8
  Week 76, n=8 | 1.0055 (33.3)
  Week 80, n=8: number analyzed (Participants) | 8
  Week 80, n=8 | 1.0431 (21.6)
  Week 84, n=8: number analyzed (Participants) | 8
  Week 84, n=8 | 0.9959 (25.3)
  Week 88, n=8: number analyzed (Participants) | 8
  Week 88, n=8 | 1.0529 (16.3)
  Week 92, n=8: number analyzed (Participants) | 8
  Week 92, n=8 | 1.0052 (26.3)
  Week 96, n=8: number analyzed (Participants) | 8
  Week 96, n=8 | 1.1204 (22.1)
  Week 100, n=8: number analyzed (Participants) | 8
  Week 100, n=8 | 1.1122 (24.7)
  Week 104, n=10: number analyzed (Participants) | 10
  Week 104, n=10 | 1.0480 (23.3)
  Week 116; n= 8: number analyzed (Participants) | 8
  Week 116; n= 8 | 1.0373 (19.8)
  Week 128, n=9: number analyzed (Participants) | 9
  Week 128, n=9 | 0.9971 (35.2)

15. Secondary Outcome: Serum Creatinine Levels at the Indicated Time Points
Description: Serum creatinine was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum creatinine is defined as the mean of the Screening and Day 0 values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micromoles/liter (µmol/L)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
micromoles/liter (µmol/L)
  Baseline; n= 14 | 97.1658 (22.8)
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 100.6421 (26.8)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 99.9535 (24.8)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 96.6583 (30.2)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 103.0265 (32.8)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 92.4547 (29.6)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 97.7260 (29.7)

16. Secondary Outcome: Change From Baseline in Serum Creatinine Levels at the Indicated Time Points
Description: Serum creatinine was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum creatinine is defined as the mean of the Screening and Day 0 values and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 1.0530 (14.8)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 1.0202 (18.6)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 1.0581 (23.7)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 0.9818 (28.7)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 0.9467 (20.1)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 0.9874 (30.4)

17. Secondary Outcome: Serum Albumin Levels at Indicated Time Points
Description: Serum albumin was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum albumin is defined as the mean of the Screening and Day 0 values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up.
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams per liter (g/L)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
grams per liter (g/L)
  Baseline; n= 14 | 23.3306 (22.7)
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 24.4204 (27.5)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 27.8397 (23.4)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 31.9927 (18.3)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 33.9484 (10.9)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 39.1015 (7.5)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 39.2009 (8.8)

18. Secondary Outcome: Change From Baseline in Levels of Serum Albumin at the Indicated Time Points
Description: Serum albumin was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum albumin is defined as the mean of the Screening and Day 0 values and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
ratio
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 1.0324 (15.0)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 1.1211 (16.9)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 1.2828 (28.1)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 1.3695 (23.8)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 1.5879 (19.6)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 1.5799 (24.7)

19. Secondary Outcome: Serum Cholesterol Levels at Indicated Time Points
Description: Serum cholesterol was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum cholesterol is defined as the mean of the Screening and Day 0 values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles per liter (mmol/L)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
millimoles per liter (mmol/L)
  Baseline; n= 14 | 7.6423 (36.0)
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 7.2336 (31.5)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 6.2740 (23.1)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 5.8724 (18.6)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 5.0211 (18.4)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 4.8001 (24.5)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 4.2407 (12.7)

20. Secondary Outcome: Change From Baseline in Serum Cholesterol at the Indicated Time Points
Description: Serum cholesterol was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum cholesterol is defined as the mean of the Screening and Day 0 values and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
mmol/L
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 0.9238 (16.8)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 0.8896 (14.3)
  Week 52; n= 7: number analyzed (Participants) | 7
  Week 52; n= 7 | 0.8571 (16.7)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 0.7111 (15.0)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 0.6851 (17.3)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 0.6140 (15.7)

21. Secondary Outcome: Serum Immunoglobulin G (IgG) Levels at Indicated Time Points
Description: Serum IgG was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum IgG is defined as the pre-dose Day 0 value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow-up
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
g/L
  Baseline; n= 14 | 4.026 (1.6810)
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 3.871 (1.5266)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 4.405 (1.7833)
  Week 52; n= 8: number analyzed (Participants) | 8
  Week 52; n= 8 | 5.823 (2.2572)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 6.050 (2.1103)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 7.611 (2.8301)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 8.609 (2.2597)

22. Secondary Outcome: Change From Baseline in Serum IgG at the Indicated Time Points
Description: Serum IgG was assessed as a clinical chemistry laboratory parameter from Baseline up to Week 128/6 month follow-up visit. Baseline for serum IgG is defined as the pre-dose Day 0 value and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, 104 and 128/6 month follow up
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  Week 12; n= 13: number analyzed (Participants) | 13
  Week 12; n= 13 | 0.055 (0.6625)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 0.469 (1.4287)
  Week 52; n= 8: number analyzed (Participants) | 8
  Week 52; n= 8 | 1.525 (2.4411)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 1.619 (1.6681)
  Week 104; n= 10: number analyzed (Participants) | 10
  Week 104; n= 10 | 3.613 (2.5488)
  Week 128; n= 9: number analyzed (Participants) | 9
  Week 128; n= 9 | 4.334 (2.0289)

23. Secondary Outcome: Number of Participants With Edema and Edema Extending Beyond Calf
Description: Reduction of proteinuria lessens the risk of thromboembolic and cardiovascular effects and reduces the edema in participants. Investigators physically reviewed participants for clinical manifestations of idiopathic membranous glomerulonephropathy (IMGN) (e.g. edema extending beyond calf) during study and analysis was performed at Week 12, 28, 52, 76 Week 104. Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Baseline and Weeks 12, 28, 52, 76, and 104
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Week 0; oedema; n= 14 | 13
  Week 0; oedema extending beyond calf; n= 14 | 5
  Week 12; oedema; n= 12 | 9
  Week 12; Oedema extending beyond calf; n= 12 | 1
  Week 28;Oedema; n= 11 | 7
  Week 28; Oedema extending beyond calf; n= 11 | 1
  Week 52; oedema; n= 9 | 4
  Week 52;Oedema extending beyond calf; n= 9 | 1
  Week 76;Oedema; n=8 | 4
  Week 76;Oedema extending beyond calf; n= 8 | 0
  4 Week post final dose (PFD); Oedema; n=10 | 6
  4 Week PFD; Oedema extending beyond calf; n= 10 | 1
  Week 104 withdrawn (WD); Oedema; n= 1 | 0
  Week 104 WD;Oedema extending beyond calf; n= 1 | 0

24. Secondary Outcome: Summary of Maximum Observed Serum Concentration (Cmax) of Belimumab at the Indicated Time Points
Description: The first occurrence of Cmax was determined directly from the serum concentration-time data. The pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis and all calculations of non-compartmental parameters are being based on actual sampling times.
Time Frame: Baseline and up to 4 week post last dose
Population: PK Population: all participants in the ITT Population for whom a PK sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
nanograms per milliliter (ng/mL)
  Day 0, 5 minutes; n= 13: number analyzed (Participants) | 13
  Day 0, 5 minutes; n= 13 | 267996.0 (70598.02)
  Week 28, 5 minutes; n= 11: number analyzed (Participants) | 11
  Week 28, 5 minutes; n= 11 | 312462.2 (95171.16)

25. Secondary Outcome: Summary of Minimum Observed Concentration (Cmin) of Belimumab at the Indicated Time Points
Description: Trough concentration (Cmin) samples collected on the specified days are being used to assess attainment whether there was sufficient belimumab despite it being lost in the urine from the proteinuria and to check if it improved as proteinuria resolved. Analysis was performed on pre-infusion samples at weeks 2,4,8,12,28,40,52,76 and the 4 week post last-dose.
Time Frame: Baseline and up to 4 week post last dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
ng/mL
  Pre-infusion; Week 2; n= 14 | 29940.8 (20918.28)
  Pre-infusion; Week 4; n= 12: number analyzed (Participants) | 12
  Pre-infusion; Week 4; n= 12 | 41220.9 (35720.14)
  Pre-infusion; Week 8; n= 13: number analyzed (Participants) | 13
  Pre-infusion; Week 8; n= 13 | 30350.9 (25505.70)
  Pre-infusion; Week 12; n= 11: number analyzed (Participants) | 11
  Pre-infusion; Week 12; n= 11 | 30913.7 (30681.42)
  Pre-infusion; Week 28; n= 11: number analyzed (Participants) | 11
  Pre-infusion; Week 28; n= 11 | 34904.7 (26388.60)
  Pre-infusion; Week 40; n= 10: number analyzed (Participants) | 10
  Pre-infusion; Week 40; n= 10 | 40800.6 (28847.86)
  Pre-infusion; Week 52; n= 9: number analyzed (Participants) | 9
  Pre-infusion; Week 52; n= 9 | 38375.9 (14136.23)
  Pre-infusion; Week 76; n= 8: number analyzed (Participants) | 8
  Pre-infusion; Week 76; n= 8 | 65655.8 (32873.33)
  4 Weeks post last-dose; n= 9: number analyzed (Participants) | 9
  4 Weeks post last-dose; n= 9 | 60497.3 (28074.37)

26. Secondary Outcome: Summary of Area Under the Serum Concentration-time Curve to the Last Quantifiable Concentration (AUC[0-2])
Description: The AUC(0-2) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples for PK analysis were collected at the following time points: pre-dose (on dosing days): Days 0, 1, 4, 7, 14 and Week 4, 8, 12, 28, 40, 52, 76 and 4 week post last dose. Post-dose (5 minutes after dosing complete): Days 0 and 28. The results will be posted at later date following post hoc analysis.
Time Frame: Baseline and up to 4 week post last dose
Population: PK Population
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0

27. Secondary Outcome: Summary of Total Amount of Urine Excreted Ae(0-24)
Description: PK parameters from the urine concentration data: urine Ae(0-24) were assessed. 24 h urine collections for PK analysis were collected after the Day 0 and Weeks 12, 28, 52, 76 doses and at the 4 week post last dose visit. A population approach was undertaken to characterize the population PK parameters and associated variability of belimumab in nephrotic participants. The population approach could have provided derived clearance of belimumab for each participant after the first dose. The population PK analysis was conducted using nonlinear mixed-effect modeling (NONMEM) or appropriate nonlinear mixed-effect analysis software. Several samples were taken pre-dose at Day 0 and some at week 12 incorrectly which affects interpretation.
Time Frame: Baseline and Up to 4 week post last dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/hour
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
ng/hour
  Day 0; n= 14 | 105826.23 (178943.857)
  Week 12; n= 12: number analyzed (Participants) | 12
  Week 12; n= 12 | 95188.14 (130217.976)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 92997.94 (110142.599)
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | 219367.96 (391752.377)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | 145645.34 (267292.225)
  4 Week post last dose; n= 6: number analyzed (Participants) | 6
  4 Week post last dose; n= 6 | 7909.34 (16771.559)

28. Secondary Outcome: Change From Baseline in Short Form (SF)-36 v2 Quality of Life (QoL) Questionnaire Score
Description: Health-related quality of life was assessed through participant self-completion of the short form health survey (SF-36 version [v2]), a general health related quality of life metrics. Norm-based Scores (NBS) for physical functioning, role emotional, role physical were assessed. The remaining SF-36 component scores require re-scaling and therefore will be added at a later date. SF-36 was administered prior to any procedures at Weeks 12, 28, 52, 76 and 104/4 week post last dose. Item score were recorded and higher score represented better health status. Baseline is defined as Day 0 pre dose value and change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Only those participants available at the specified time points were analyzed (represented by n=X in category titles).
Time Frame: Baseline and up to Week 104/4 week post last dose
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Scores on a scale
  Physical functioning, Week 12; n= 12: number analyzed (Participants) | 12
  Physical functioning, Week 12; n= 12 | -4.034 (5.1907)
  Physical functioning, Week 28; n= 11: number analyzed (Participants) | 11
  Physical functioning, Week 28; n= 11 | -0.765 (3.6780)
  Physical functioning, Week 52; n= 9: number analyzed (Participants) | 9
  Physical functioning, Week 52; n= 9 | 0.468 (7.3489)
  Physical functioning, Week 76; n= 7: number analyzed (Participants) | 7
  Physical functioning, Week 76; n= 7 | 0.601 (7.9409)
  Physical functioning 4 Week post final dose;n=11: number analyzed (Participants) | 11
  Physical functioning 4 Week post final dose;n=11 | 0.765 (11.7275)
  Role emotional, Week 12; n= 12: number analyzed (Participants) | 12
  Role emotional, Week 12; n= 12 | -0.000 (10.4831)
  Role emotional, Week 28; n= 11: number analyzed (Participants) | 11
  Role emotional, Week 28; n= 11 | 1.413 (15.1824)
  Role emotional, Week 52; n= 9: number analyzed (Participants) | 9
  Role emotional, Week 52; n= 9 | 3.023 (11.4621)
  Role emotional, Week 76; n= 7: number analyzed (Participants) | 7
  Role emotional, Week 76; n= 7 | 3.332 (7.2475)
  Role emotional, 4 Week post final dose; n= 11: number analyzed (Participants) | 11
  Role emotional, 4 Week post final dose; n= 11 | 6.007 (10.0413)
  Role physical, Week 12; n= 12: number analyzed (Participants) | 12
  Role physical, Week 12; n= 12 | 0.816 (11.0681)
  Role physical, Week 28; n= 11: number analyzed (Participants) | 11
  Role physical, Week 28; n= 11 | 3.340 (8.4324)
  Role physical, Week 52; n= 9: number analyzed (Participants) | 9
  Role physical, Week 52; n= 9 | 3.537 (9.1726)
  Role physical, Week 76; n= 7: number analyzed (Participants) | 7
  Role physical, Week 76; n= 7 | 7.697 (12.2803)
  Role physical 4 Week post final dose; n= 11: number analyzed (Participants) | 11
  Role physical 4 Week post final dose; n= 11 | 5.789 (11.4489)

29. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The analysis was performed on Safety Population which comprised of all participants who were randomized into the study. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, Requires hospitalization or prolongation of existing hospitalization, Results in disability/incapacity, is a congenital anomaly/birth defect, may require medical or surgical intervention, is associated with liver injury and impaired liver function.
Time Frame: Baseline and up to Week 128/6 month follow up
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  AE | 14
  SAE | 3

30. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry and Hematology Values
Description: Blood samples were collected from participants for evaluation of clinical chemistry and hematology parameters. The clinical chemistry parameters included albumin, alkaline phosphatase (alk.phosph.), alanine amino transferase (ALT), aspartate amino transferase (AST), total and direct bilirubin, calcium, cholesterol, chloride, carbon dioxide, creatinine, gamma glutamyl transferase (GGT), glucose, potassium, lactate dehydrogenase (LD), magnesium, sodium, phosphorus, total protein, blood urea nitrogen (BUN) and uric acid. The hematology parameters included basophils, eosinophil, hemoglobin, hematocrit, lymphocytes, monocytes, total neutrophils, platelets, red blood cells (RBC) count and white blood cells (WBC) count. Participants were counted in the category that their value changes to (low or high) for the specific time points. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 116/16 week follow-up visit
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Albumin; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Albumin; Week 12; to high; n= 13 | 0
  Albumin; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Albumin; Week 12; to low; n= 13 | 0
  Albumin; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Albumin; Week 28; to high; n= 11 | 0
  Albumin; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Albumin; Week 28; to low; n= 11 | 0
  Albumin; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Albumin; Week 52; to high; n= 7 | 0
  Albumin; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Albumin; Week 52; to low; n= 7 | 0
  Albumin; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Albumin; Week 76; to high; n= 8 | 0
  Albumin; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Albumin; Week 76; to low; n= 8 | 0
  Albumin; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Albumin; Week 104; to high; n= 10 | 0
  Albumin; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Albumin; Week 104; to low; n= 10 | 0
  Albumin; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Albumin; 16 Week follow up; to high; n= 8 | 0
  Albumin; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Albumin; 16 Week follow up; to low; n= 8 | 0
  Alk.phosph.; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Alk.phosph.; Week 12; to high; n= 13 | 0
  Alk.phosph.; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Alk.phosph.; Week 12; to low; n= 13 | 0
  Alk.phosph.; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Alk.phosph.; Week 28; to high; n= 11 | 0
  Alk.phosph.; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Alk.phosph.; Week 28; to low; n= 11 | 0
  Alk.phosph.; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Alk.phosph.; Week 52; to high; n= 7 | 0
  Alk.phosph.; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Alk.phosph.; Week 52; to low; n= 7 | 0
  Alk.phosph.; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Alk.phosph.; Week 76; to high; n= 8 | 0
  Alk.phosph.; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Alk.phosph.; Week 76; to low; n= 8 | 0
  Alk.phosph.; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Alk.phosph.; Week 104; to high; n= 10 | 0
  Alk.phosph.; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Alk.phosph.; Week 104; to low; n= 10 | 0
  Alk.phosph.; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Alk.phosph.; 16 Week follow up; to high; n= 8 | 0
  Alk.phosph.; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Alk.phosph.; 16 Week follow up; to low; n= 8 | 0
  ALT; Week 12; to high; n= 13: number analyzed (Participants) | 13
  ALT; Week 12; to high; n= 13 | 0
  ALT; Week 12; to low; n= 13: number analyzed (Participants) | 13
  ALT; Week 12; to low; n= 13 | 0
  ALT; Week 28; to high; n= 11: number analyzed (Participants) | 11
  ALT; Week 28; to high; n= 11 | 0
  ALT; Week 28; to low; n= 11: number analyzed (Participants) | 11
  ALT; Week 28; to low; n= 11 | 0
  ALT; Week 52; to high; n= 7: number analyzed (Participants) | 7
  ALT; Week 52; to high; n= 7 | 0
  ALT; Week 52; to low; n= 7: number analyzed (Participants) | 7
  ALT; Week 52; to low; n= 7 | 0
  ALT; Week 76; to high; n= 8: number analyzed (Participants) | 8
  ALT; Week 76; to high; n= 8 | 0
  ALT; Week 76; to low; n= 8: number analyzed (Participants) | 8
  ALT; Week 76; to low; n= 8 | 0
  ALT; Week 104; to high; n= 10: number analyzed (Participants) | 10
  ALT; Week 104; to high; n= 10 | 0
  ALT; Week 104; to low; n= 10: number analyzed (Participants) | 10
  ALT; Week 104; to low; n= 10 | 0
  ALT; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  ALT; 16 Week follow up; to high; n= 8 | 0
  ALT; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  ALT; 16 Week follow up; to low; n= 8 | 0
  AST; Week 12; to high; n= 13: number analyzed (Participants) | 13
  AST; Week 12; to high; n= 13 | 0
  AST; Week 12; to low; n= 13: number analyzed (Participants) | 13
  AST; Week 12; to low; n= 13 | 0
  AST; Week 28; to high; n= 11: number analyzed (Participants) | 11
  AST; Week 28; to high; n= 11 | 1
  AST; Week 28; to low; n= 11: number analyzed (Participants) | 11
  AST; Week 28; to low; n= 11 | 0
  AST; Week 52; to high; n= 7: number analyzed (Participants) | 7
  AST; Week 52; to high; n= 7 | 0
  AST; Week 52; to low; n= 7: number analyzed (Participants) | 7
  AST; Week 52; to low; n= 7 | 0
  AST; Week 76; to high; n= 8: number analyzed (Participants) | 8
  AST; Week 76; to high; n= 8 | 0
  AST; Week 76; to low; n= 8: number analyzed (Participants) | 8
  AST; Week 76; to low; n= 8 | 0
  AST; Week 104; to high; n= 10: number analyzed (Participants) | 10
  AST; Week 104; to high; n= 10 | 0
  AST; Week 104; to low; n= 10: number analyzed (Participants) | 10
  AST; Week 104; to low; n= 10 | 0
  AST; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  AST; 16 Week follow up; to high; n= 8 | 0
  AST; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  AST; 16 Week follow up; to low; n= 8 | 0
  Direct bilirubin; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Direct bilirubin; Week 12; to high; n= 13 | 0
  Direct bilirubin; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Direct bilirubin; Week 12; to low; n= 13 | 0
  Direct bilirubin; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Direct bilirubin; Week 28; to high; n= 11 | 0
  Direct bilirubin; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Direct bilirubin; Week 28; to low; n= 11 | 0
  Direct bilirubin; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Direct bilirubin; Week 52; to high; n= 7 | 0
  Direct bilirubin; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Direct bilirubin; Week 52; to low; n= 7 | 0
  Direct bilirubin; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Direct bilirubin; Week 76; to high; n= 8 | 0
  Direct bilirubin; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Direct bilirubin; Week 76; to low; n= 8 | 0
  Direct bilirubin; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Direct bilirubin; Week 104; to high; n= 10 | 0
  Direct bilirubin; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Direct bilirubin; Week 104; to low; n= 10 | 0
  Direct bilirubin; 16 Week follow up; to high; n=8: number analyzed (Participants) | 8
  Direct bilirubin; 16 Week follow up; to high; n=8 | 0
  Direct bilirubin; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Direct bilirubin; 16 Week follow up; to low; n= 8 | 0
  Total bilirubin; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Total bilirubin; Week 12; to high; n= 12 | 0
  Total bilirubin; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Total bilirubin; Week 12; to low; n= 12 | 0
  Total bilirubin; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Total bilirubin; Week 28; to high; n= 11 | 0
  Total bilirubin; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Total bilirubin; Week 28; to low; n= 11 | 0
  Total bilirubin; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Total bilirubin; Week 52; to high; n= 7 | 0
  Total bilirubin; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Total bilirubin; Week 52; to low; n= 7 | 0
  Total bilirubin; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Total bilirubin; Week 76; to high; n= 8 | 0
  Total bilirubin; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Total bilirubin; Week 76; to low; n= 8 | 0
  Total bilirubin; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Total bilirubin; Week 104; to high; n= 10 | 0
  Total bilirubin; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Total bilirubin; Week 104; to low; n= 10 | 0
  Total bilirubin; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Total bilirubin; 16 Week follow up; to high; n= 8 | 0
  Total bilirubin; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Total bilirubin; 16 Week follow up; to low; n= 8 | 0
  Calcium; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Calcium; Week 12; to high; n= 12 | 0
  Calcium; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Calcium; Week 12; to low; n= 12 | 0
  Calcium; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Calcium; Week 28; to high; n= 11 | 0
  Calcium; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Calcium; Week 28; to low; n= 11 | 0
  Calcium; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Calcium; Week 52; to high; n= 7 | 0
  Calcium; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Calcium; Week 52; to low; n= 7 | 0
  Calcium; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Calcium; Week 76; to high; n= 8 | 0
  Calcium; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Calcium; Week 76; to low; n= 8 | 0
  Calcium; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Calcium; Week 104; to high; n= 10 | 1
  Calcium; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Calcium; Week 104; to low; n= 10 | 1
  Calcium; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Calcium; 16 Week follow up; to high; n= 8 | 0
  Calcium; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Calcium; 16 Week follow up; to low; n= 8 | 0
  Cholesterol; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Cholesterol; Week 12; to high; n= 13 | 0
  Cholesterol; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Cholesterol; Week 12; to low; n= 13 | 0
  Cholesterol; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Cholesterol; Week 28; to high; n= 11 | 0
  Cholesterol; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Cholesterol; Week 28; to low; n= 11 | 0
  Cholesterol; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Cholesterol; Week 52; to high; n= 7 | 0
  Cholesterol; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Cholesterol; Week 52; to low; n= 7 | 0
  Cholesterol; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Cholesterol; Week 76; to high; n= 8 | 0
  Cholesterol; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Cholesterol; Week 76; to low; n= 8 | 0
  Cholesterol; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Cholesterol; Week 104; to high; n= 10 | 0
  Cholesterol; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Cholesterol; Week 104; to low; n= 10 | 0
  Cholesterol; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Cholesterol; 16 Week follow up; to high; n= 8 | 0
  Cholesterol; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Cholesterol; 16 Week follow up; to low; n= 8 | 0
  Chloride; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Chloride; Week 12; to high; n= 13 | 1
  Chloride; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Chloride; Week 12; to low; n= 13 | 0
  Chloride; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Chloride; Week 28; to high; n= 11 | 2
  Chloride; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Chloride; Week 28; to low; n= 11 | 0
  Chloride; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Chloride; Week 52; to high; n= 7 | 0
  Chloride; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Chloride; Week 52; to low; n= 7 | 0
  Chloride; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Chloride; Week 76; to high; n= 8 | 0
  Chloride; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Chloride; Week 76; to low; n= 8 | 0
  Chloride; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Chloride; Week 104; to high; n= 10 | 0
  Chloride; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Chloride; Week 104; to low; n= 10 | 0
  Chloride; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Chloride; 16 Week follow up; to high; n= 8 | 0
  Chloride; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Chloride; 16 Week follow up; to low; n= 8 | 0
  Carbon dioxide; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Carbon dioxide; Week 12; to high; n= 13 | 0
  Carbon dioxide; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Carbon dioxide; Week 12; to low; n= 13 | 1
  Carbon dioxide; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Carbon dioxide; Week 28; to high; n= 11 | 0
  Carbon dioxide; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Carbon dioxide; Week 28; to low; n= 11 | 3
  Carbon dioxide; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Carbon dioxide; Week 52; to high; n= 7 | 0
  Carbon dioxide; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Carbon dioxide; Week 52; to low; n= 7 | 0
  Carbon dioxide; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Carbon dioxide; Week 76; to high; n= 8 | 0
  Carbon dioxide; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Carbon dioxide; Week 76; to low; n= 8 | 0
  Carbon dioxide; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Carbon dioxide; Week 104; to high; n= 10 | 0
  Carbon dioxide; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Carbon dioxide; Week 104; to low; n= 10 | 1
  Carbon dioxide; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Carbon dioxide; 16 Week follow up; to high; n= 8 | 0
  Carbon dioxide; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Carbon dioxide; 16 Week follow up; to low; n= 8 | 0
  Creatinine; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Creatinine; Week 12; to high; n= 13 | 2
  Creatinine; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Creatinine; Week 12; to low; n= 13 | 0
  Creatinine; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Creatinine; Week 28; to high; n= 11 | 0
  Creatinine; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Creatinine; Week 28; to low; n= 11 | 0
  Creatinine; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Creatinine; Week 52; to high; n= 7 | 0
  Creatinine; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Creatinine; Week 52; to low; n= 7 | 0
  Creatinine; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Creatinine; Week 76; to high; n= 8 | 2
  Creatinine; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Creatinine; Week 76; to low; n= 8 | 1
  Creatinine; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Creatinine; Week 104; to high; n= 10 | 0
  Creatinine; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Creatinine; Week 104; to low; n= 10 | 0
  Creatinine; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Creatinine; 16 Week follow up; to high; n= 8 | 0
  Creatinine; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Creatinine; 16 Week follow up; to low; n= 8 | 0
  GGT; Week 12; to high; n= 13: number analyzed (Participants) | 13
  GGT; Week 12; to high; n= 13 | 0
  GGT; Week 12; to low; n= 13: number analyzed (Participants) | 13
  GGT; Week 12; to low; n= 13 | 0
  GGT; Week 28; to high; n= 11: number analyzed (Participants) | 11
  GGT; Week 28; to high; n= 11 | 0
  GGT; Week 28; to low; n= 11: number analyzed (Participants) | 11
  GGT; Week 28; to low; n= 11 | 0
  GGT; Week 52; to high; n= 7: number analyzed (Participants) | 7
  GGT; Week 52; to high; n= 7 | 0
  GGT; Week 52; to low; n= 7: number analyzed (Participants) | 7
  GGT; Week 52; to low; n= 7 | 0
  GGT; Week 76; to high; n= 8: number analyzed (Participants) | 8
  GGT; Week 76; to high; n= 8 | 0
  GGT; Week 76; to low; n= 8: number analyzed (Participants) | 8
  GGT; Week 76; to low; n= 8 | 0
  GGT; Week 104; to high; n= 10: number analyzed (Participants) | 10
  GGT; Week 104; to high; n= 10 | 0
  GGT; Week 104; to low; n= 10: number analyzed (Participants) | 10
  GGT; Week 104; to low; n= 10 | 0
  GGT; 16 Week follow up; to high; n=8: number analyzed (Participants) | 8
  GGT; 16 Week follow up; to high; n=8 | 0
  GGT; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  GGT; 16 Week follow up; to low; n= 8 | 0
  Glucose; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Glucose; Week 12; to high; n= 13 | 3
  Glucose; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Glucose; Week 12; to low; n= 13 | 0
  Glucose; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Glucose; Week 28; to high; n= 11 | 4
  Glucose; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Glucose; Week 28; to low; n= 11 | 0
  Glucose; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Glucose; Week 52; to high; n= 7 | 2
  Glucose; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Glucose; Week 52; to low; n= 7 | 0
  Glucose; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Glucose; Week 76; to high; n= 8 | 3
  Glucose; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Glucose; Week 76; to low; n= 8 | 0
  Glucose; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Glucose; Week 104; to high; n= 10 | 1
  Glucose; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Glucose; Week 104; to low; n= 10 | 0
  Glucose; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Glucose; 16 Week follow up; to high; n= 8 | 1
  Glucose; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Glucose; 16 Week follow up; to low; n= 8 | 1
  Potassium; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Potassium; Week 12; to high; n= 13 | 0
  Potassium; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Potassium; Week 12; to low; n= 13 | 0
  Potassium; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Potassium; Week 28; to high; n= 11 | 1
  Potassium; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Potassium; Week 28; to low; n= 11 | 1
  Potassium; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Potassium; Week 52; to high; n= 7 | 0
  Potassium; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Potassium; Week 52; to low; n= 7 | 0
  Potassium; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Potassium; Week 76; to high; n= 8 | 0
  Potassium; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Potassium; Week 76; to low; n= 8 | 0
  Potassium; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Potassium; Week 104; to high; n= 10 | 0
  Potassium; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Potassium; Week 104; to low; n= 10 | 0
  Potassium; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Potassium; 16 Week follow up; to high; n= 8 | 0
  Potassium; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Potassium; 16 Week follow up; to low; n= 8 | 0
  LD; Week 12; to high; n= 13: number analyzed (Participants) | 13
  LD; Week 12; to high; n= 13 | 3
  LD; Week 12; to low; n= 13: number analyzed (Participants) | 13
  LD; Week 12; to low; n= 13 | 0
  LD; Week 28; to high; n= 11: number analyzed (Participants) | 11
  LD; Week 28; to high; n= 11 | 2
  LD; Week 28; to low; n= 11: number analyzed (Participants) | 11
  LD; Week 28; to low; n= 11 | 0
  LD; Week 52; to high; n= 7: number analyzed (Participants) | 7
  LD; Week 52; to high; n= 7 | 1
  LD; Week 52; to low; n= 7: number analyzed (Participants) | 7
  LD; Week 52; to low; n= 7 | 0
  LD; Week 76; to high; n= 8: number analyzed (Participants) | 8
  LD; Week 76; to high; n= 8 | 1
  LD; Week 76; to low; n= 8: number analyzed (Participants) | 8
  LD; Week 76; to low; n= 8 | 0
  LD;Week 104; to high; n= 10: number analyzed (Participants) | 10
  LD;Week 104; to high; n= 10 | 0
  LD;Week 104; to low; n= 10: number analyzed (Participants) | 10
  LD;Week 104; to low; n= 10 | 0
  LD; 16 week follow-up; to high; n= 8: number analyzed (Participants) | 8
  LD; 16 week follow-up; to high; n= 8 | 0
  LD; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  LD; 16 week follow up; to low; n= 8 | 0
  Magnesium; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Magnesium; Week 12; to high; n= 13 | 1
  Magnesium; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Magnesium; Week 12; to low; n= 13 | 0
  Magnesium; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Magnesium; Week 28; to high; n= 11 | 0
  Magnesium; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Magnesium; Week 28; to low; n= 11 | 0
  Magnesium; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Magnesium; Week 52; to high; n= 7 | 0
  Magnesium; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Magnesium; Week 52; to low; n= 7 | 0
  Magnesium; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Magnesium; Week 76; to high; n= 8 | 0
  Magnesium; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Magnesium; Week 76; to low; n= 8 | 0
  Magnesium; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Magnesium; Week 104; to high; n= 10 | 0
  Magnesium; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Magnesium; Week 104; to low; n= 10 | 0
  Magnesium; 16 week follow up; to high; n= 8: number analyzed (Participants) | 8
  Magnesium; 16 week follow up; to high; n= 8 | 0
  Magnesium; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  Magnesium; 16 week follow up; to low; n= 8 | 0
  Sodium; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Sodium; Week 12; to high; n= 12 | 0
  Sodium; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Sodium; Week 12; to low; n= 12 | 0
  Sodium; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Sodium; Week 28; to high; n= 11 | 0
  Sodium; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Sodium; Week 28; to low; n= 11 | 1
  Sodium; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Sodium; Week 52; to high; n= 7 | 0
  Sodium; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Sodium; Week 52; to low; n= 7 | 1
  Sodium; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Sodium; Week 76; to high; n= 8 | 0
  Sodium; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Sodium; Week 76; to low; n= 8 | 1
  Sodium; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Sodium; Week 104; to high; n= 10 | 0
  Sodium; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Sodium; Week 104; to low; n= 10 | 0
  Sodium; 16 week follow p; to high; n= 8: number analyzed (Participants) | 8
  Sodium; 16 week follow p; to high; n= 8 | 0
  Sodium; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  Sodium; 16 week follow up; to low; n= 8 | 1
  Phosphorus; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Phosphorus; Week 12; to high; n= 13 | 1
  Phosphorus; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Phosphorus; Week 12; to low; n= 13 | 0
  Phosphorus; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Phosphorus; Week 28; to high; n= 11 | 2
  Phosphorus; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Phosphorus; Week 28; to low; n= 11 | 0
  Phosphorus; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Phosphorus; Week 52; to high; n= 7 | 0
  Phosphorus; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Phosphorus; Week 52; to low; n= 7 | 0
  Phosphorus; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Phosphorus; Week 76; to high; n= 8 | 0
  Phosphorus; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Phosphorus; Week 76; to low; n= 8 | 0
  Phosphorus;Week 104; to high; n= 10: number analyzed (Participants) | 10
  Phosphorus;Week 104; to high; n= 10 | 1
  Phosphorus;Week 104; to low; n= 10: number analyzed (Participants) | 10
  Phosphorus;Week 104; to low; n= 10 | 1
  Phosphorus; 16 week follow up; to high; n= 8: number analyzed (Participants) | 8
  Phosphorus; 16 week follow up; to high; n= 8 | 0
  Phosphorus; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  Phosphorus; 16 week follow up; to low; n= 8 | 0
  Total protein; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Total protein; Week 12; to high; n= 12 | 0
  Total protein; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Total protein; Week 12; to low; n= 12 | 0
  Total protein; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Total protein; Week 28; to high; n= 11 | 0
  Total protein; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Total protein; Week 28; to low; n= 11 | 0
  Total protein; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Total protein; Week 52; to high; n= 7 | 0
  Total protein; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Total protein; Week 52; to low; n= 7 | 1
  Total protein; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Total protein; Week 76; to high; n= 8 | 0
  Total protein; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Total protein; Week 76; to low; n= 8 | 0
  Total protein; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Total protein; Week 104; to high; n= 10 | 0
  Total protein; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Total protein; Week 104; to low; n= 10 | 0
  Total protein; 16 Week follow up; to high; n= 8: number analyzed (Participants) | 8
  Total protein; 16 Week follow up; to high; n= 8 | 0
  Total protein; 16 Week follow up; to low; n= 8: number analyzed (Participants) | 8
  Total protein; 16 Week follow up; to low; n= 8 | 0
  BUN; Week 12; to high; n= 13: number analyzed (Participants) | 13
  BUN; Week 12; to high; n= 13 | 2
  BUN; Week 12; to low; n= 13: number analyzed (Participants) | 13
  BUN; Week 12; to low; n= 13 | 0
  BUN; Week 28; to high; n= 11: number analyzed (Participants) | 11
  BUN; Week 28; to high; n= 11 | 0
  BUN; Week 28; to low; n= 11: number analyzed (Participants) | 11
  BUN; Week 28; to low; n= 11 | 0
  BUN; Week 52; to high; n= 7: number analyzed (Participants) | 7
  BUN; Week 52; to high; n= 7 | 2
  BUN; Week 52; to low; n= 7: number analyzed (Participants) | 7
  BUN; Week 52; to low; n= 7 | 0
  BUN; Week 76; to high; n= 8: number analyzed (Participants) | 8
  BUN; Week 76; to high; n= 8 | 2
  BUN; Week 76; to low; n= 8: number analyzed (Participants) | 8
  BUN; Week 76; to low; n= 8 | 0
  BUN; Week 104; to high; n= 10: number analyzed (Participants) | 10
  BUN; Week 104; to high; n= 10 | 0
  BUN; Week 104; to low; n= 10: number analyzed (Participants) | 10
  BUN; Week 104; to low; n= 10 | 0
  BUN; 16 week follow up; to high; n= 8: number analyzed (Participants) | 8
  BUN; 16 week follow up; to high; n= 8 | 0
  BUN; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  BUN; 16 week follow up; to low; n= 8 | 0
  Uric acid; Week 12; to high; n= 13: number analyzed (Participants) | 13
  Uric acid; Week 12; to high; n= 13 | 2
  Uric acid; Week 12; to low; n= 13: number analyzed (Participants) | 13
  Uric acid; Week 12; to low; n= 13 | 2
  Uric acid; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Uric acid; Week 28; to high; n= 11 | 1
  Uric acid; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Uric acid; Week 28; to low; n= 11 | 0
  Uric acid; Week 52; to high; n= 7: number analyzed (Participants) | 7
  Uric acid; Week 52; to high; n= 7 | 1
  Uric acid; Week 52; to low; n= 7: number analyzed (Participants) | 7
  Uric acid; Week 52; to low; n= 7 | 0
  Uric acid; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Uric acid; Week 76; to high; n= 8 | 2
  Uric acid; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Uric acid; Week 76; to low; n= 8 | 0
  Uric acid; Week 104; to high; n= 10: number analyzed (Participants) | 10
  Uric acid; Week 104; to high; n= 10 | 2
  Uric acid; Week 104; to low; n= 10: number analyzed (Participants) | 10
  Uric acid; Week 104; to low; n= 10 | 0
  Uric acid; 16 week follow up; to high; n= 8: number analyzed (Participants) | 8
  Uric acid; 16 week follow up; to high; n= 8 | 2
  Uric acid; 16 week follow up; to low; n= 8: number analyzed (Participants) | 8
  Uric acid; 16 week follow up; to low; n= 8 | 0
  Basophils; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Basophils; Week 12; to high; n= 12 | 0
  Basophils; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Basophils; Week 12; to low; n= 12 | 0
  Basophils; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Basophils; Week 28; to high; n= 11 | 0
  Basophils; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Basophils; Week 28; to low; n= 11 | 0
  Basophils; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Basophils; Week 52; to high; n= 9 | 0
  Basophils; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Basophils; Week 52; to low; n= 9 | 0
  Basophils; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Basophils; Week 76; to high; n= 8 | 0
  Basophils; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Basophils; Week 76; to low; n= 8 | 0
  Basophils; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Basophils; Week 104; to high; n= 9 | 0
  Basophils; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Basophils; Week 104; to low; n= 9 | 0
  Basophils; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Basophils; 16 week follow up; to high; n= 9 | 0
  Basophils; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Basophils; 16 week follow up; to low; n= 9 | 0
  Eosinophils; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Eosinophils; Week 12; to high; n= 12 | 1
  Eosinophils; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Eosinophils; Week 12; to low; n= 12 | 0
  Eosinophils; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Eosinophils; Week 28; to high; n= 11 | 1
  Eosinophils; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Eosinophils; Week 28; to low; n= 11 | 0
  Eosinophils; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Eosinophils; Week 52; to high; n= 9 | 0
  Eosinophils; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Eosinophils; Week 52; to low; n= 9 | 0
  Eosinophils; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Eosinophils; Week 76; to high; n= 8 | 1
  Eosinophils; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Eosinophils; Week 76; to low; n= 8 | 0
  Eosinophils; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Eosinophils; Week 104; to high; n= 9 | 0
  Eosinophils; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Eosinophils; Week 104; to low; n= 9 | 0
  Eosinophils; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Eosinophils; 16 week follow up; to high; n= 9 | 0
  Eosinophils; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Eosinophils; 16 week follow up; to low; n= 9 | 0
  Hemoglobin; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Hemoglobin; Week 12; to high; n= 12 | 0
  Hemoglobin; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Hemoglobin; Week 12; to low; n= 12 | 0
  Hemoglobin; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Hemoglobin; Week 28; to high; n= 11 | 0
  Hemoglobin; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Hemoglobin; Week 28; to low; n= 11 | 0
  Hemoglobin; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Hemoglobin; Week 52; to high; n= 9 | 0
  Hemoglobin; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Hemoglobin; Week 52; to low; n= 9 | 2
  Hemoglobin; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Hemoglobin; Week 76; to high; n= 8 | 0
  Hemoglobin; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Hemoglobin; Week 76; to low; n= 8 | 1
  Hemoglobin; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Hemoglobin; Week 104; to high; n= 9 | 0
  Hemoglobin; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Hemoglobin; Week 104; to low; n= 9 | 1
  Hemoglobin; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Hemoglobin; 16 week follow up; to high; n= 9 | 0
  Hemoglobin; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Hemoglobin; 16 week follow up; to low; n= 9 | 1
  Hematocrit; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Hematocrit; Week 12; to high; n= 12 | 0
  Hematocrit; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Hematocrit; Week 12; to low; n= 12 | 0
  Hematocrit; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Hematocrit; Week 28; to high; n= 11 | 1
  Hematocrit; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Hematocrit; Week 28; to low; n= 11 | 0
  Hematocrit; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Hematocrit; Week 52; to high; n= 9 | 0
  Hematocrit; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Hematocrit; Week 52; to low; n= 9 | 1
  Hematocrit; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Hematocrit; Week 76; to high; n= 8 | 0
  Hematocrit; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Hematocrit; Week 76; to low; n= 8 | 0
  Hematocrit; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Hematocrit; Week 104; to high; n= 9 | 0
  Hematocrit; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Hematocrit; Week 104; to low; n= 9 | 1
  Hematocrit; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Hematocrit; 16 week follow up; to high; n= 9 | 0
  Hematocrit; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Hematocrit; 16 week follow up; to low; n= 9 | 1
  Lymphocytes; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Lymphocytes; Week 12; to high; n= 12 | 0
  Lymphocytes; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Lymphocytes; Week 12; to low; n= 12 | 0
  Lymphocytes; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Lymphocytes; Week 28; to high; n= 11 | 0
  Lymphocytes; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Lymphocytes; Week 28; to low; n= 11 | 0
  Lymphocytes; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Lymphocytes; Week 52; to high; n= 9 | 0
  Lymphocytes; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Lymphocytes; Week 52; to low; n= 9 | 0
  Lymphocytes; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Lymphocytes; Week 76; to high; n= 8 | 0
  Lymphocytes; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Lymphocytes; Week 76; to low; n= 8 | 0
  Lymphocytes; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Lymphocytes; Week 104; to high; n= 9 | 0
  Lymphocytes; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Lymphocytes; Week 104; to low; n= 9 | 0
  Lymphocytes; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Lymphocytes; 16 week follow up; to high; n= 9 | 0
  Lymphocytes; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Lymphocytes; 16 week follow up; to low; n= 9 | 0
  Monocytes; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Monocytes; Week 12; to high; n= 12 | 0
  Monocytes; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Monocytes; Week 12; to low; n= 12 | 0
  Monocytes; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Monocytes; Week 28; to high; n= 11 | 0
  Monocytes; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Monocytes; Week 28; to low; n= 11 | 0
  Monocytes; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Monocytes; Week 52; to high; n= 9 | 0
  Monocytes; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Monocytes; Week 52; to low; n= 9 | 0
  Monocytes; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Monocytes; Week 76; to high; n= 8 | 0
  Monocytes; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Monocytes; Week 76; to low; n= 8 | 0
  Monocytes; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Monocytes; Week 104; to high; n= 9 | 0
  Monocytes; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Monocytes; Week 104; to low; n= 9 | 0
  Monocytes; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Monocytes; 16 week follow up; to high; n= 9 | 0
  Monocytes; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Monocytes; 16 week follow up; to low; n= 9 | 0
  Neutrophils; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Neutrophils; Week 12; to high; n= 12 | 1
  Neutrophils; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Neutrophils; Week 12; to low; n= 12 | 0
  Neutrophils; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Neutrophils; Week 28; to high; n= 11 | 0
  Neutrophils; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Neutrophils; Week 28; to low; n= 11 | 0
  Neutrophils; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Neutrophils; Week 52; to high; n= 9 | 0
  Neutrophils; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Neutrophils; Week 52; to low; n= 9 | 0
  Neutrophils; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Neutrophils; Week 76; to high; n= 8 | 0
  Neutrophils; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Neutrophils; Week 76; to low; n= 8 | 0
  Neutrophils; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Neutrophils; Week 104; to high; n= 9 | 2
  Neutrophils; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Neutrophils; Week 104; to low; n= 9 | 0
  Neutrophils; 16 week follow up; to high; n=9: number analyzed (Participants) | 9
  Neutrophils; 16 week follow up; to high; n=9 | 1
  Neutrophils; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Neutrophils; 16 week follow up; to low; n= 9 | 0
  Platelet count; Week 12; to high; n= 12: number analyzed (Participants) | 12
  Platelet count; Week 12; to high; n= 12 | 3
  Platelet count; Week 12; to low; n= 12: number analyzed (Participants) | 12
  Platelet count; Week 12; to low; n= 12 | 0
  Platelet count; Week 28; to high; n= 11: number analyzed (Participants) | 11
  Platelet count; Week 28; to high; n= 11 | 2
  Platelet count; Week 28; to low; n= 11: number analyzed (Participants) | 11
  Platelet count; Week 28; to low; n= 11 | 0
  Platelet count; Week 52; to high; n= 9: number analyzed (Participants) | 9
  Platelet count; Week 52; to high; n= 9 | 0
  Platelet count; Week 52; to low; n= 9: number analyzed (Participants) | 9
  Platelet count; Week 52; to low; n= 9 | 0
  Platelet count; Week 76; to high; n= 8: number analyzed (Participants) | 8
  Platelet count; Week 76; to high; n= 8 | 0
  Platelet count; Week 76; to low; n= 8: number analyzed (Participants) | 8
  Platelet count; Week 76; to low; n= 8 | 0
  Platelet count; Week 104; to high; n= 9: number analyzed (Participants) | 9
  Platelet count; Week 104; to high; n= 9 | 1
  Platelet count; Week 104; to low; n= 9: number analyzed (Participants) | 9
  Platelet count; Week 104; to low; n= 9 | 0
  Platelet count; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  Platelet count; 16 week follow up; to high; n= 9 | 0
  Platelet count; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  Platelet count; 16 week follow up; to low; n= 9 | 0
  RBC; Week 12; to high; n= 12: number analyzed (Participants) | 12
  RBC; Week 12; to high; n= 12 | 0
  RBC; Week 12; to low; n= 12: number analyzed (Participants) | 12
  RBC; Week 12; to low; n= 12 | 3
  RBC; Week 28; to high; n= 11: number analyzed (Participants) | 11
  RBC; Week 28; to high; n= 11 | 0
  RBC; Week 28; to low; n= 11: number analyzed (Participants) | 11
  RBC; Week 28; to low; n= 11 | 1
  RBC; Week 52; to high; n= 9: number analyzed (Participants) | 9
  RBC; Week 52; to high; n= 9 | 0
  RBC; Week 52; to low; n= 9: number analyzed (Participants) | 9
  RBC; Week 52; to low; n= 9 | 1
  RBC; Week 76; to high; n= 8: number analyzed (Participants) | 8
  RBC; Week 76; to high; n= 8 | 0
  RBC; Week 76; to low; n= 8: number analyzed (Participants) | 8
  RBC; Week 76; to low; n= 8 | 0
  RBC; Week 104; to high; n= 9: number analyzed (Participants) | 9
  RBC; Week 104; to high; n= 9 | 0
  RBC; Week 104; to low; n= 9: number analyzed (Participants) | 9
  RBC; Week 104; to low; n= 9 | 0
  RBC; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  RBC; 16 week follow up; to high; n= 9 | 0
  RBC; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  RBC; 16 week follow up; to low; n= 9 | 1
  WBC; Week 12; to high; n= 12: number analyzed (Participants) | 12
  WBC; Week 12; to high; n= 12 | 1
  WBC; Week 12; to low; n= 12: number analyzed (Participants) | 12
  WBC; Week 12; to low; n= 12 | 0
  WBC; Week 28; to high; n= 11: number analyzed (Participants) | 11
  WBC; Week 28; to high; n= 11 | 0
  WBC; Week 28; to low; n= 11: number analyzed (Participants) | 11
  WBC; Week 28; to low; n= 11 | 0
  WBC; Week 52; to high; n= 9: number analyzed (Participants) | 9
  WBC; Week 52; to high; n= 9 | 0
  WBC; Week 52; to low; n= 9: number analyzed (Participants) | 9
  WBC; Week 52; to low; n= 9 | 0
  WBC; Week 76; to high; n= 8: number analyzed (Participants) | 8
  WBC; Week 76; to high; n= 8 | 0
  WBC; Week 76; to low; n= 8: number analyzed (Participants) | 8
  WBC; Week 76; to low; n= 8 | 0
  WBC; Week 104; to high; n= 9: number analyzed (Participants) | 9
  WBC; Week 104; to high; n= 9 | 2
  WBC; Week 104; to low; n= 9: number analyzed (Participants) | 9
  WBC; Week 104; to low; n= 9 | 0
  WBC; 16 week follow up; to high; n= 9: number analyzed (Participants) | 9
  WBC; 16 week follow up; to high; n= 9 | 1
  WBC; 16 week follow up; to low; n= 9: number analyzed (Participants) | 9
  WBC; 16 week follow up; to low; n= 9 | 0

31. Secondary Outcome: Number of Participants With Urinalysis Dipstick Findings
Description: Urine samples were collected for urinalysis by dipstick method from Baseline up to Week 116/16 months follow up and number of participants with findings were presented for Baseline, Week 12, 28, 52, 76, 104/4 weeks post last-dose and Week 116/16 week follow up (WF). The urinalysis parameters included occult blood, glucose, ketones, protein. The findings were presented as trace or 1/10 g/100 milliliter (dL), trace, negative, 4+, 3+, 3+ or 1 g/dL, 2+ or 1/2 g/dL, 2+, 1+ or 1/4 g/dL and 1+. Only participants present at the specific time points were presented (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 116/16 Week follow up
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants
  Week 12; occult blood; Trace or 1/10 g/DL; n= 12: number analyzed (Participants) | 12
  Week 12; occult blood; Trace or 1/10 g/DL; n= 12 | 0
  Week 12;Occult Blood; Trace; n= 12: number analyzed (Participants) | 12
  Week 12;Occult Blood; Trace; n= 12 | 1
  Week 12; Occult Blood; negative; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; negative; n= 12 | 2
  Week 12; Occult Blood; 4+; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 4+; n= 12 | 0
  Week 12; Occult Blood; 3+ OR 1 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 3+ OR 1 G/DL; n= 12 | 0
  Week 12; Occult Blood; 3+; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 3+; n= 12 | 2
  Week 12; Occult Blood; 2+ OR 1/2 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 2+ OR 1/2 G/DL; n= 12 | 0
  Week 12; Occult Blood; 2+ ; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 2+ ; n= 12 | 6
  Week 12; Occult Blood;1+ OR 1/4 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood;1+ OR 1/4 G/DL; n= 12 | 0
  Week 12; Occult Blood; 1+; n= 12: number analyzed (Participants) | 12
  Week 12; Occult Blood; 1+; n= 12 | 1
  Week 12; glucose; Trace or 1/10 g/DL; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; Trace or 1/10 g/DL; n= 12 | 3
  Week 12;glucose; Trace; n= 12: number analyzed (Participants) | 12
  Week 12;glucose; Trace; n= 12 | 0
  Week 12; glucose; negative; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; negative; n= 12 | 8
  Week 12; glucose; 4+; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 4+; n= 12 | 0
  Week 12; glucose; 3+ OR 1 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 3+ OR 1 G/DL; n= 12 | 0
  Week 12; glucose; 3+; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 3+; n= 12 | 0
  Week 12; glucose; 2+ OR 1/2 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 2+ OR 1/2 G/DL; n= 12 | 0
  Week 12; glucose; 2+ ; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 2+ ; n= 12 | 0
  Week 12; glucose;1+ OR 1/4 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; glucose;1+ OR 1/4 G/DL; n= 12 | 1
  Week 12; glucose; 1+; n= 12: number analyzed (Participants) | 12
  Week 12; glucose; 1+; n= 12 | 0
  Week 12; ketones; Trace or 1/10 g/DL; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; Trace or 1/10 g/DL; n= 12 | 0
  Week 12; ketones; Trace; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; Trace; n= 12 | 0
  Week 12; ketones; negative; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; negative; n= 12 | 12
  Week 12; ketones; 4+; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 4+; n= 12 | 0
  Week 12; ketones; 3+ OR 1 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 3+ OR 1 G/DL; n= 12 | 0
  Week 12; ketones; 3+; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 3+; n= 12 | 0
  Week 12; ketones; 2+ OR 1/2 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 2+ OR 1/2 G/DL; n= 12 | 0
  Week 12; ketones; 2+ ; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 2+ ; n= 12 | 0
  Week 12; ketones;1+ OR 1/4 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; ketones;1+ OR 1/4 G/DL; n= 12 | 0
  Week 12; ketones; 1+; n= 12: number analyzed (Participants) | 12
  Week 12; ketones; 1+; n= 12 | 0
  Week 12; protein; Trace or 1/10 g/DL; n= 12: number analyzed (Participants) | 12
  Week 12; protein; Trace or 1/10 g/DL; n= 12 | 0
  Week 12; Protein; Trace; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; Trace; n= 12 | 0
  Week 12; Protein; negative; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; negative; n= 12 | 0
  Week 12; Protein; 4+; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 4+; n= 12 | 0
  Week 12; Protein; 3+ OR 1 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 3+ OR 1 G/DL; n= 12 | 0
  Week 12; Protein; 3+; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 3+; n= 12 | 8
  Week 12; Protein; 2+ OR 1/2 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 2+ OR 1/2 G/DL; n= 12 | 0
  Week 12; Protein; 2+ ; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 2+ ; n= 12 | 3
  Week 12; Protein;1+ OR 1/4 G/DL; n= 12: number analyzed (Participants) | 12
  Week 12; Protein;1+ OR 1/4 G/DL; n= 12 | 0
  Week 12; Protein; 1+; n= 12: number analyzed (Participants) | 12
  Week 12; Protein; 1+; n= 12 | 1
  Week 28; occult blood; Trace or 1/10 g/DL; n= 11: number analyzed (Participants) | 11
  Week 28; occult blood; Trace or 1/10 g/DL; n= 11 | 0
  Week 28;Occult Blood; Trace; n= 11: number analyzed (Participants) | 11
  Week 28;Occult Blood; Trace; n= 11 | 2
  Week 28; Occult Blood; negative; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; negative; n= 11 | 1
  Week 28; Occult Blood; 4+; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 4+; n= 11 | 0
  Week 28; Occult Blood; 3+ OR 1 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 3+ OR 1 G/DL; n= 11 | 0
  Week 28; Occult Blood; 3+; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 3+; n= 11 | 0
  Week 28; Occult Blood; 2+ OR 1/2 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 2+ OR 1/2 G/DL; n= 11 | 0
  Week 28; Occult Blood; 2+ ; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 2+ ; n= 11 | 4
  Week 28; Occult Blood;1+ OR 1/4 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood;1+ OR 1/4 G/DL; n= 11 | 0
  Week 28; Occult Blood; 1+; n= 11: number analyzed (Participants) | 11
  Week 28; Occult Blood; 1+; n= 11 | 4
  Week 28; glucose; Trace or 1/10 g/DL; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; Trace or 1/10 g/DL; n= 11 | 1
  Week 28;glucose; Trace; n= 11: number analyzed (Participants) | 11
  Week 28;glucose; Trace; n= 11 | 0
  Week 28; glucose; negative; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; negative; n= 11 | 9
  Week 28; glucose; 4+; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 4+; n= 11 | 0
  Week 28; glucose; 3+ OR 1 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 3+ OR 1 G/DL; n= 11 | 0
  Week 28; glucose; 3+; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 3+; n= 11 | 0
  Week 28; glucose; 2+ OR 1/2 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 2+ OR 1/2 G/DL; n= 11 | 0
  Week 28; glucose; 2+ ; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 2+ ; n= 11 | 0
  Week 28; glucose;1+ OR 1/4 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; glucose;1+ OR 1/4 G/DL; n= 11 | 1
  Week 28; glucose; 1+; n= 11: number analyzed (Participants) | 11
  Week 28; glucose; 1+; n= 11 | 0
  Week 28; ketones; Trace or 1/10 g/DL; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; Trace or 1/10 g/DL; n= 11 | 0
  Week 28; ketones; Trace; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; Trace; n= 11 | 0
  Week 28; ketones; negative; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; negative; n= 11 | 11
  Week 28; ketones; 4+; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 4+; n= 11 | 0
  Week 28; ketones; 3+ OR 1 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 3+ OR 1 G/DL; n= 11 | 0
  Week 28; ketones; 3+; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 3+; n= 11 | 0
  Week 28; ketones; 2+ OR 1/2 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 2+ OR 1/2 G/DL; n= 11 | 0
  Week 28; ketones; 2+ ; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 2+ ; n= 11 | 0
  Week 28; ketones;1+ OR 1/4 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; ketones;1+ OR 1/4 G/DL; n= 11 | 0
  Week 28; ketones; 1+; n= 11: number analyzed (Participants) | 11
  Week 28; ketones; 1+; n= 11 | 0
  Week 28; protein; Trace or 1/10 g/DL; n= 11: number analyzed (Participants) | 11
  Week 28; protein; Trace or 1/10 g/DL; n= 11 | 0
  Week 28; Protein; Trace; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; Trace; n= 11 | 0
  Week 28; Protein; negative; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; negative; n= 11 | 0
  Week 28; protein; 4+; n= 11: number analyzed (Participants) | 11
  Week 28; protein; 4+; n= 11 | 0
  Week 28; Protein; 3+ OR 1 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; 3+ OR 1 G/DL; n= 11 | 0
  Week 28; Protein; 3+; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; 3+; n= 11 | 10
  Week 28; Protein; 2+ OR 1/2 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; 2+ OR 1/2 G/DL; n= 11 | 0
  Week 28; Protein; 2+ ; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; 2+ ; n= 11 | 1
  Week 28; Protein;1+ OR 1/4 G/DL; n= 11: number analyzed (Participants) | 11
  Week 28; Protein;1+ OR 1/4 G/DL; n= 11 | 0
  Week 28; Protein; 1+; n= 11: number analyzed (Participants) | 11
  Week 28; Protein; 1+; n= 11 | 0
  Week 52; occult blood; Trace or 1/10 g/DL; n= 9: number analyzed (Participants) | 9
  Week 52; occult blood; Trace or 1/10 g/DL; n= 9 | 0
  Week 52;Occult Blood; Trace; n= 9: number analyzed (Participants) | 9
  Week 52;Occult Blood; Trace; n= 9 | 2
  Week 52; Occult Blood; negative; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; negative; n= 9 | 3
  Week 52; Occult Blood; 4+; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 4+; n= 9 | 0
  Week 52; Occult Blood; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 3+ OR 1 G/DL; n= 9 | 0
  Week 52; Occult Blood; 3+; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 3+; n= 9 | 0
  Week 52; Occult Blood; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 2+ OR 1/2 G/DL; n= 9 | 0
  Week 52; Occult Blood; 2+ ; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 2+ ; n= 9 | 4
  Week 52; Occult Blood;1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood;1+ OR 1/4 G/DL; n= 9 | 0
  Week 52; Occult Blood; 1+; n= 9: number analyzed (Participants) | 9
  Week 52; Occult Blood; 1+; n= 9 | 0
  Week 52; glucose; Trace or 1/10 g/DL; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; Trace or 1/10 g/DL; n= 9 | 2
  Week 52;glucose; Trace; n= 9: number analyzed (Participants) | 9
  Week 52;glucose; Trace; n= 9 | 0
  Week 52; glucose; negative; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; negative; n= 9 | 7
  Week 52; glucose; 4+; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 4+; n= 9 | 0
  Week 52; glucose; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 3+ OR 1 G/DL; n= 9 | 0
  Week 52; glucose; 3+; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 3+; n= 9 | 0
  Week 52; glucose; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 2+ OR 1/2 G/DL; n= 9 | 0
  Week 52; glucose; 2+ ; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 2+ ; n= 9 | 0
  Week 52; glucose;1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; glucose;1+ OR 1/4 G/DL; n= 9 | 0
  Week 52; glucose; 1+; n= 9: number analyzed (Participants) | 9
  Week 52; glucose; 1+; n= 9 | 0
  Week 52; ketones; Trace or 1/10 g/DL; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; Trace or 1/10 g/DL; n= 9 | 0
  Week 52; ketones; Trace; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; Trace; n= 9 | 0
  Week 52; ketones; negative; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; negative; n= 9 | 9
  Week 52; ketones; 4+; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 4+; n= 9 | 0
  Week 52; ketones; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 3+ OR 1 G/DL; n= 9 | 0
  Week 52; ketones; 3+; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 3+; n= 9 | 0
  Week 52; ketones; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 2+ OR 1/2 G/DL; n= 9 | 0
  Week 52; ketones; 2+ ; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 2+ ; n= 9 | 0
  Week 52; ketones;1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; ketones;1+ OR 1/4 G/DL; n= 9 | 0
  Week 52; ketones; 1+; n= 9: number analyzed (Participants) | 9
  Week 52; ketones; 1+; n= 9 | 0
  Week 52; protein; Trace or 1/10 g/DL; n= 9: number analyzed (Participants) | 9
  Week 52; protein; Trace or 1/10 g/DL; n= 9 | 0
  Week 52; Protein; Trace; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; Trace; n= 9 | 0
  Week 52; Protein; negative; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; negative; n= 9 | 0
  Week 52; protein; 4+; n= 9: number analyzed (Participants) | 9
  Week 52; protein; 4+; n= 9 | 0
  Week 52; Protein; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; 3+ OR 1 G/DL; n= 9 | 0
  Week 52; Protein; 3+; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; 3+; n= 9 | 4
  Week 52; Protein; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; 2+ OR 1/2 G/DL; n= 9 | 0
  Week 52; Protein; 2+ ; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; 2+ ; n= 9 | 3
  Week 52; Protein;1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  Week 52; Protein;1+ OR 1/4 G/DL; n= 9 | 0
  Week 52; Protein; 1+; n= 9: number analyzed (Participants) | 9
  Week 52; Protein; 1+; n= 9 | 2
  Week 76; occult blood; Trace or 1/10 g/DL;n=7: number analyzed (Participants) | 7
  Week 76; occult blood; Trace or 1/10 g/DL;n=7 | 0
  Week 76;Occult Blood; Trace; n= 7: number analyzed (Participants) | 7
  Week 76;Occult Blood; Trace; n= 7 | 3
  Week 76; Occult Blood; negative; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; negative; n= 7 | 3
  Week 76; Occult Blood; 4+; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 4+; n= 7 | 0
  Week 76; Occult Blood; 3+ OR 1 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 3+ OR 1 G/DL; n= 7 | 0
  Week 76; Occult Blood; 3+; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 3+; n= 7 | 0
  Week 76; Occult Blood; 2+ OR 1/2 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 2+ OR 1/2 G/DL; n= 7 | 0
  Week 76; Occult Blood; 2+ ; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 2+ ; n= 7 | 0
  Week 76; Occult Blood;1+ OR 1/4 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood;1+ OR 1/4 G/DL; n= 7 | 0
  Week 76; Occult Blood; 1+; n= 7: number analyzed (Participants) | 7
  Week 76; Occult Blood; 1+; n= 7 | 1
  Week 76; glucose; Trace or 1/10 g/DL; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; Trace or 1/10 g/DL; n= 7 | 2
  Week 76;glucose; Trace; n= 7: number analyzed (Participants) | 7
  Week 76;glucose; Trace; n= 7 | 0
  Week 76; glucose; negative; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; negative; n= 7 | 5
  Week 76; glucose; 4+; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 4+; n= 7 | 0
  Week 76; glucose; 3+ OR 1 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 3+ OR 1 G/DL; n= 7 | 0
  Week 76; glucose; 3+; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 3+; n= 7 | 0
  Week 76; glucose; 2+ OR 1/2 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 2+ OR 1/2 G/DL; n= 7 | 0
  Week 76; glucose; 2+ ; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 2+ ; n= 7 | 0
  Week 76; glucose;1+ OR 1/4 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; glucose;1+ OR 1/4 G/DL; n= 7 | 0
  Week 76; glucose; 1+; n= 7: number analyzed (Participants) | 7
  Week 76; glucose; 1+; n= 7 | 0
  Week 76; ketones; Trace or 1/10 g/DL; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; Trace or 1/10 g/DL; n= 7 | 0
  Week 76; ketones; Trace; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; Trace; n= 7 | 0
  Week 76; ketones; negative; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; negative; n= 7 | 7
  Week 76; ketones; 4+; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 4+; n= 7 | 0
  Week 76; ketones; 3+ OR 1 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 3+ OR 1 G/DL; n= 7 | 0
  Week 76; ketones; 3+; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 3+; n= 7 | 0
  Week 76; ketones; 2+ OR 1/2 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 2+ OR 1/2 G/DL; n= 7 | 0
  Week 76; ketones; 2+ ; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 2+ ; n= 7 | 0
  Week 76; ketones;1+ OR 1/4 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; ketones;1+ OR 1/4 G/DL; n= 7 | 0
  Week 76; ketones; 1+; n= 7: number analyzed (Participants) | 7
  Week 76; ketones; 1+; n= 7 | 0
  Week 76; protein; Trace or 1/10 g/DL; n= 7: number analyzed (Participants) | 7
  Week 76; protein; Trace or 1/10 g/DL; n= 7 | 0
  Week 76; Protein; Trace; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; Trace; n= 7 | 0
  Week 76; Protein; negative; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; negative; n= 7 | 1
  Week 76; protein; 4+; n= 7: number analyzed (Participants) | 7
  Week 76; protein; 4+; n= 7 | 0
  Week 76; Protein; 3+ OR 1 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; 3+ OR 1 G/DL; n= 7 | 0
  Week 76; Protein; 3+; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; 3+; n= 7 | 1
  Week 76; Protein; 2+ OR 1/2 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; 2+ OR 1/2 G/DL; n= 7 | 0
  Week 76; Protein; 2+ ; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; 2+ ; n= 7 | 4
  Week 76; Protein;1+ OR 1/4 G/DL; n= 7: number analyzed (Participants) | 7
  Week 76; Protein;1+ OR 1/4 G/DL; n= 7 | 0
  Week 76; Protein; 1+; n= 7: number analyzed (Participants) | 7
  Week 76; Protein; 1+; n= 7 | 1
  Week 104; occult blood; Trace or 1/10 g/DL;n=10: number analyzed (Participants) | 10
  Week 104; occult blood; Trace or 1/10 g/DL;n=10 | 0
  Week 104;Occult Blood; Trace; n= 10: number analyzed (Participants) | 10
  Week 104;Occult Blood; Trace; n= 10 | 0
  Week 104; Occult Blood; negative; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; negative; n= 10 | 8
  Week 104; Occult Blood; 4+; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 4+; n= 10 | 0
  Week 104; Occult Blood; 3+ OR 1 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 3+ OR 1 G/DL; n= 10 | 0
  Week 104; Occult Blood; 3+; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 3+; n= 10 | 0
  Week 104; Occult Blood; 2+ OR 1/2 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 2+ OR 1/2 G/DL; n= 10 | 0
  Week 104; Occult Blood; 2+ ; n=10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 2+ ; n=10 | 1
  Week 104; Occult Blood;1+ OR 1/4 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood;1+ OR 1/4 G/DL; n= 10 | 0
  Week 104; Occult Blood; 1+; n= 10: number analyzed (Participants) | 10
  Week 104; Occult Blood; 1+; n= 10 | 1
  Week 104; glucose; Trace or 1/10 g/DL; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; Trace or 1/10 g/DL; n= 10 | 2
  Week 104 ;glucose; Trace; n= 10: number analyzed (Participants) | 10
  Week 104 ;glucose; Trace; n= 10 | 0
  Week 104; glucose; negative; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; negative; n= 10 | 7
  Week 104; glucose; 4+; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 4+; n= 10 | 0
  Week 104; glucose; 3+ OR 1 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 3+ OR 1 G/DL; n= 10 | 0
  Week 104; glucose; 3+; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 3+; n= 10 | 0
  Week 104; glucose; 2+ OR 1/2 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 2+ OR 1/2 G/DL; n= 10 | 0
  Week 104; glucose; 2+ ; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 2+ ; n= 10 | 0
  Week 104; glucose;1+ OR 1/4 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; glucose;1+ OR 1/4 G/DL; n= 10 | 1
  Week 104; glucose; 1+; n= 10: number analyzed (Participants) | 10
  Week 104; glucose; 1+; n= 10 | 0
  Week 104; ketones; Trace or 1/10 g/DL; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; Trace or 1/10 g/DL; n= 10 | 0
  Week 104; ketones; Trace; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; Trace; n= 10 | 0
  Week 104; ketones; negative; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; negative; n= 10 | 10
  Week 104; ketones; 4+; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 4+; n= 10 | 0
  Week 104; ketones; 3+ OR 1 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 3+ OR 1 G/DL; n= 10 | 0
  Week 104; ketones; 3+; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 3+; n= 10 | 0
  Week 104; ketones; 2+ OR 1/2 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 2+ OR 1/2 G/DL; n= 10 | 0
  Week 104; ketones; 2+ ; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 2+ ; n= 10 | 0
  Week 104; ketones;1+ OR 1/4 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; ketones;1+ OR 1/4 G/DL; n= 10 | 0
  Week 104; ketones; 1+; n= 10: number analyzed (Participants) | 10
  Week 104; ketones; 1+; n= 10 | 0
  Week 104; protein; Trace or 1/10 g/DL; n= 10: number analyzed (Participants) | 10
  Week 104; protein; Trace or 1/10 g/DL; n= 10 | 0
  Week 104; Protein; Trace; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; Trace; n= 10 | 0
  Week 104; Protein; negative; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; negative; n= 10 | 1
  Week 104; protein; 4+; n= 10: number analyzed (Participants) | 10
  Week 104; protein; 4+; n= 10 | 0
  Week 104; Protein; 3+ OR 1 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; 3+ OR 1 G/DL; n= 10 | 0
  Week 104; Protein; 3+; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; 3+; n= 10 | 3
  Week 104; Protein; 2+ OR 1/2 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; 2+ OR 1/2 G/DL; n= 10 | 0
  Week 104; Protein; 2+ ; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; 2+ ; n= 10 | 6
  Week 104; Protein;1+ OR 1/4 G/DL; n= 10: number analyzed (Participants) | 10
  Week 104; Protein;1+ OR 1/4 G/DL; n= 10 | 0
  Week 104; Protein; 1+; n= 10: number analyzed (Participants) | 10
  Week 104; Protein; 1+; n= 10 | 0
  16 WF; Occult blood; TRACE OR 1/10 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; TRACE OR 1/10 G/DL; n= 9 | 0
  16 WF; Occult blood; TRACE; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; TRACE; n= 9 | 2
  16 WF; Occult blood; NEGATIVE; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; NEGATIVE; n= 9 | 6
  16 WF; Occult blood; 4+; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 4+; n= 9 | 0
  16 WF; Occult blood; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 3+ OR 1 G/DL; n= 9 | 0
  16 WF; Occult blood; 3+; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 3+; n= 9 | 0
  16 WF; Occult blood; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 2+ OR 1/2 G/DL; n= 9 | 0
  16 WF; Occult blood; 2+; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 2+; n= 9 | 1
  16 WF; Occult blood; 1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 1+ OR 1/4 G/DL; n= 9 | 0
  16 WF; Occult blood; 1+; n= 9: number analyzed (Participants) | 9
  16 WF; Occult blood; 1+; n= 9 | 0
  16 WF; Glucose; TRACE OR 1/10 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; TRACE OR 1/10 G/DL; n= 9 | 1
  16 WF; Glucose; TRACE; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; TRACE; n= 9 | 0
  16 WF; Glucose; negative; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; negative; n= 9 | 7
  16 WF; Glucose; 4+; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; 4+; n= 9 | 0
  16 WF; Glucose; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; 3+ OR 1 G/DL; n= 9 | 0
  16 WF; Glucose; 3+; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; 3+; n= 9 | 0
  16 WF; Glucose; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; 2+ OR 1/2 G/DL; n= 9 | 1
  16 WF; Glucose; 2+; n= 9: number analyzed (Participants) | 9
  16 WF; Glucose; 2+; n= 9 | 0
  16 WF; Glucose; 1+ OR 1/4 G/DL; n=9: number analyzed (Participants) | 9
  16 WF; Glucose; 1+ OR 1/4 G/DL; n=9 | 0
  16 WF; Glucose; 1+; n=9: number analyzed (Participants) | 9
  16 WF; Glucose; 1+; n=9 | 0
  16 WF; Ketones; TRACE OR 1/10 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; TRACE OR 1/10 G/DL; n= 9 | 0
  16 WF; Ketones; TRACE; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; TRACE; n= 9 | 0
  16 WF; Ketones; negative; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; negative; n= 9 | 9
  16 WF; Ketones; 4+; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 4+; n= 9 | 0
  16 WF; Ketones; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 3+ OR 1 G/DL; n= 9 | 0
  16 WF; Ketones; 3+; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 3+; n= 9 | 0
  16 WF; Ketones; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 2+ OR 1/2 G/DL; n= 9 | 0
  16 WF; Ketones; 2+; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 2+; n= 9 | 0
  16 WF; Ketones; 1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 1+ OR 1/4 G/DL; n= 9 | 0
  16 WF; Ketones; 1+; n= 9: number analyzed (Participants) | 9
  16 WF; Ketones; 1+; n= 9 | 0
  16 WF; Protein; TRACE OR 1/10 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; TRACE OR 1/10 G/DL; n= 9 | 0
  16 WF; Protein; TRACE; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; TRACE; n= 9 | 1
  16 WF; Protein; negative; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; negative; n= 9 | 0
  16 WF; Protein; 4+; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 4+; n= 9 | 0
  16 WF; Protein; 3+ OR 1 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 3+ OR 1 G/DL; n= 9 | 0
  16 WF; Protein; 3+; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 3+; n= 9 | 3
  16 WF; Protein; 2+ OR 1/2 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 2+ OR 1/2 G/DL; n= 9 | 0
  16 WF; Protein; 2+; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 2+; n= 9 | 4
  16 WF; Protein; 1+ OR 1/4 G/DL; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 1+ OR 1/4 G/DL; n= 9 | 0
  16 WF; Protein; 1+; n= 9: number analyzed (Participants) | 9
  16 WF; Protein; 1+; n= 9 | 1

32. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured from Baseline throughout the treatment period up to Week 116/ 16 week follow-up visit. The Baseline value was taken at Day 0 pre dose and change from Baseline was defined as post dose visit value minus Baseline value. Mean and standard deviation (SD) were measured and presented for Week 12, 28, 52, 76, 104 withdrawn visit, 4 Week post last dose and 16 Week follow-up visit. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to week 116/16 week follow-up visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
millimeter of mercury (mmHg)
  Week 12; SBP; n= 12: number analyzed (Participants) | 12
  Week 12; SBP; n= 12 | -4.2 (17.23)
  Week 28; SBP; n= 11: number analyzed (Participants) | 11
  Week 28; SBP; n= 11 | -5.8 (18.14)
  Week 52; SBP; n= 9: number analyzed (Participants) | 9
  Week 52; SBP; n= 9 | -1.9 (18.66)
  Week 76; SBP; n= 8: number analyzed (Participants) | 8
  Week 76; SBP; n= 8 | -1.3 (11.30)
  4 Week post last dose; SBP; n= 10: number analyzed (Participants) | 10
  4 Week post last dose; SBP; n= 10 | -12.2 (11.78)
  16 Week follow up; SBP; n= 9: number analyzed (Participants) | 9
  16 Week follow up; SBP; n= 9 | -7.4 (15.72)
  Week 104 withdrawn visit; SBP; n= 2: number analyzed (Participants) | 2
  Week 104 withdrawn visit; SBP; n= 2 | -1.0 (5.66)
  Week 12; DBP; n= 12: number analyzed (Participants) | 12
  Week 12; DBP; n= 12 | 3.8 (12.94)
  Week 28; DBP; n= 11: number analyzed (Participants) | 11
  Week 28; DBP; n= 11 | 0.8 (10.75)
  Week 52; DBP; n= 9: number analyzed (Participants) | 9
  Week 52; DBP; n= 9 | 1.2 (11.87)
  Week 76; DBP; n= 8: number analyzed (Participants) | 8
  Week 76; DBP; n= 8 | 2.8 (9.68)
  4 Week post last dose; DBP; n= 10: number analyzed (Participants) | 10
  4 Week post last dose; DBP; n= 10 | -3.3 (9.87)
  16 Week follow up; DBP; n= 9: number analyzed (Participants) | 9
  16 Week follow up; DBP; n= 9 | 2.4 (14.98)
  Week 104 withdrawn visit; DBP; n= 2: number analyzed (Participants) | 2
  Week 104 withdrawn visit; DBP; n= 2 | 5.5 (2.12)

33. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured from Baseline throughout the treatment period up to Week 116/ 16 week follow-up visit. The Baseline value was taken at Day 0 pre dose and change from Baseline was defined as post dose visit value minus Baseline value. Mean and standard deviation (SD) were measured and presented for Week 12, 28, 52, 76, 104 withdrawn visit, 4 Week post last dose and 16 Week post last dose visits. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Week 116/16 week follow-up visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Beats per minute
  Week 12; n= 12: number analyzed (Participants) | 12
  Week 12; n= 12 | -0.7 (11.40)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | 1.0 (7.90)
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | -1.7 (13.11)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | -2.3 (15.77)
  4 Week post last dose; n= 10: number analyzed (Participants) | 10
  4 Week post last dose; n= 10 | -2.8 (15.33)
  16 Week follow up; n= 9: number analyzed (Participants) | 9
  16 Week follow up; n= 9 | -0.9 (16.72)
  Week 104 withdrawn visit; n= 2: number analyzed (Participants) | 2
  Week 104 withdrawn visit; n= 2 | 5.0 (7.07)

34. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured from Baseline throughout the treatment period up to Week 116/ 16 week follow-up visit. The Baseline value was taken at Day 0 pre dose and change from Baseline was defined as post dose visit value minus Baseline value. Mean and standard deviation (SD) were measured and presented for Week 12, 28, 52, 76, 104 withdrawn visit, 4 Week post last dose and 16 week post last dose visits. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Week 116/16 week follow-up visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Celsius
  Week 12; n= 12: number analyzed (Participants) | 12
  Week 12; n= 12 | -0.09 (0.591)
  Week 28; n= 11: number analyzed (Participants) | 11
  Week 28; n= 11 | -0.00 (0.453)
  Week 52; n= 9: number analyzed (Participants) | 9
  Week 52; n= 9 | -0.11 (0.639)
  Week 76; n= 8: number analyzed (Participants) | 8
  Week 76; n= 8 | -0.17 (0.486)
  4 Week post last dose; n= 8: number analyzed (Participants) | 8
  4 Week post last dose; n= 8 | -0.06 (0.604)
  16 Week follow up; n= 6: number analyzed (Participants) | 6
  16 Week follow up; n= 6 | 0.30 (0.424)
  Week 104 withdrawn visit; n= 2: number analyzed (Participants) | 2
  Week 104 withdrawn visit; n= 2 | 0.15 (0.353)

35. Secondary Outcome: Number of Participants With Positive Immunogenicity Findings
Description: Blood samples of participants were collected pre-dose on Weeks 0, 12, 28, 40, 52, 76, 4 week post last dose and 16 week post last dose visit for belimumab immunogenicity assay. No participants showed positive immunogenicity findings.
Time Frame: Baseline and up to Week 116/16 week follow-up visit
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Participants | 0

36. Secondary Outcome: Urine Membrane Attack Complex (MAC) Levels
Description: Urine membrane attack complex was assayed quantitatively by ELISA method. Urine MAC samples were collected at Day 0 and Weeks 8, 28, 52, 76 and 4 week post last dose. Results were normalized using urine creatinine concentration to adjust for urine dilution. Endpoint was moved to 'Exploratory' in Protocol amendment 5 as risk of availability of functioning assay for urine membrane attack complex was noted. No assay was subsequently found and samples were not analyzed
Time Frame: Baseline and up to 4 week post last dose
Population: ITT Population
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0

37. Secondary Outcome: Change From Baseline in Urine Membrane Attack Complex (MAC)
Description: Urine membrane attack complex will be assayed quantitatively by ELISA method. Urine MAC samples are being collected at Day 0 and Weeks 8, 28, 52, 76 and 4 week post last dose. Results will be normalized using urine creatinine concentration to adjust for urine dilution, before calculation of the ratio as value at time point divided by value at Baseline (Day 0). Endpoint was changed to 'exploratory' as risk of availability of functioning assay for urine membrane attack complex was noted. No assay was subsequently found and samples were not analyzed.
Time Frame: Baseline and up to 4 week post last dose
Population: ITT Population
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0

38. Secondary Outcome: Change From Baseline in B Cell and T Cell Markers Concentration
Description: B cell Facs panels were used to measure changes over the course of therapy in B cell subsets such as transitional, naïve, memory and plasma B cell compartments by percent of the B cell compartments and absolute numbers. T cell Facs panel were used to measure changes in T cell subsets, such as T regs and CD4+ and CD8+ T cells, in terms of numbers and expression of activation markers to establish if B cell targeting with belimumab affects the T cell compartment perhaps through limiting B cell antigen presentation or cytokine release. Baseline is defined as Day 0 value and change from Baseline was calculated as ratio of post-Baseline value divided by the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 128/6 month post last dose
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
Ratio
  CD19+; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+; Week 8; n= 12 | 0.7221 (82.1)
  CD19+; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+; Week 16; n= 11 | 0.9209 (63.6)
  CD19+; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+; Week 28; n= 10 | 1.0049 (71.6)
  CD19+; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+; Week 104; n= 10 | 0.5193 (156.2)
  CD19+; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+; 6 month follow up; n= 7 | 0.3828 (185.7)
  CD19+ CD24b+ CD38b+ CD27-; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+ CD24b+ CD38b+ CD27-; Week 8; n= 12 | 0.2352 (340.0)
  CD19+ CD24b+ CD38b+ CD27-; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+ CD24b+ CD38b+ CD27-; Week 16; n= 11 | 0.6228 (316.7)
  CD19+ CD24b+ CD38b+ CD27-; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+ CD24b+ CD38b+ CD27-; Week 28; n= 10 | 0.6119 (656.0)
  CD19+ CD24b+ CD38b+ CD27-; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+ CD24b+ CD38b+ CD27-; Week 104; n= 10 | 0.3582 (405.1)
  CD19+ CD24b+ CD38b+ CD27-; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+ CD24b+ CD38b+ CD27-; 6 month follow up; n= 7 | 1.6471 (534.0)
  CD19+ CD27- IgD+; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+ CD27- IgD+; Week 8; n= 12 | 0.3490 (131.6)
  CD19+ CD27- IgD+; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+ CD27- IgD+; Week 16; n= 11 | 0.4486 (94.7)
  CD19+ CD27- IgD+; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+ CD27- IgD+; Week 28; n= 10 | 0.4561 (82.5)
  CD19+ CD27- IgD+; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+ CD27- IgD+; Week 104; n= 10 | 0.1808 (298.6)
  CD19+ CD27- IgD+; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+ CD27- IgD+; 6 month follow up; n= 7 | 0.3278 (189.2)
  CD19+ CD27-; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+ CD27-; Week 8; n= 12 | 0.4074 (109.2)
  CD19+ CD27-; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+ CD27-; Week 16; n= 11 | 0.5079 (88.1)
  CD19+ CD27-; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+ CD27-; Week 28; n= 10 | 0.5165 (76.5)
  CD19+ CD27-; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+ CD27-; Week 104; n= 10 | 0.2602 (236.9)
  CD19+ CD27-; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+ CD27-; 6 month follow up; n= 7 | 0.3756 (186.0)
  CD19lo CD38hi CD27hi; Week 8; n= 12: number analyzed (Participants) | 12
  CD19lo CD38hi CD27hi; Week 8; n= 12 | 0.5982 (555.4)
  CD19lo CD38hi CD27hi; Week 16; n= 11: number analyzed (Participants) | 11
  CD19lo CD38hi CD27hi; Week 16; n= 11 | 0.4128 (1085.7)
  CD19lo CD38hi CD27hi; Week 28; n= 10: number analyzed (Participants) | 10
  CD19lo CD38hi CD27hi; Week 28; n= 10 | 0.4481 (651.6)
  CD19lo CD38hi CD27hi; Week 104; n= 10: number analyzed (Participants) | 10
  CD19lo CD38hi CD27hi; Week 104; n= 10 | 0.2615 (238.8)
  CD19lo CD38hi CD27hi; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19lo CD38hi CD27hi; 6 month follow up; n= 7 | 0.0647 (1269.7)
  CD19+ CD24+ CD27+ ; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+ CD24+ CD27+ ; Week 8; n= 12 | 2.0747 (65.3)
  CD19+ CD24+ CD27+ ; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+ CD24+ CD27+ ; Week 16; n= 11 | 2.4161 (61.2)
  CD19+ CD24+ CD27+ ; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+ CD24+ CD27+ ; Week 28; n= 10 | 3.1294 (64.2)
  CD19+ CD24+ CD27+ ; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+ CD24+ CD27+ ; Week 104; n= 10 | 0.6089 (104014.8)
  CD19+ CD24+ CD27+ ; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+ CD24+ CD27+ ; 6 month follow up; n= 7 | 0.7952 (328.6)
  CD19+CD27+; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+CD27+; Week 8; n= 12 | 1.9195 (69.9)
  CD19+CD27+; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+CD27+; Week 16; n= 11 | 2.3132 (62.7)
  CD19+CD27+; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+CD27+; Week 28; n= 10 | 3.1352 (65.6)
  CD19+CD27+; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+CD27+; Week 104; n= 10 | 1.3273 (127.7)
  CD19+CD27+; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+CD27+; 6 month follow up; n= 7 | 0.3338 (158.2)
  CD19+CD27+IgD; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+CD27+IgD; Week 8; n= 12 | 1.9365 (69.6)
  CD19+CD27+IgD; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+CD27+IgD; Week 16; n= 11 | 2.3147 (75.1)
  CD19+CD27+IgD; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+CD27+IgD; Week 28; n= 10 | 3.2313 (51.1)
  CD19+CD27+IgD; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+CD27+IgD; Week 104; n= 10 | 1.2814 (102.3)
  CD19+CD27+IgD; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+CD27+IgD; 6 month follow up; n= 7 | 0.2413 (163.9)
  CD19+CD27+IgD-; Week 8; n= 12: number analyzed (Participants) | 12
  CD19+CD27+IgD-; Week 8; n= 12 | 1.8846 (67.7)
  CD19+CD27+IgD-; Week 16; n= 11: number analyzed (Participants) | 11
  CD19+CD27+IgD-; Week 16; n= 11 | 2.2113 (70.4)
  CD19+CD27+IgD-; Week 28; n= 10: number analyzed (Participants) | 10
  CD19+CD27+IgD-; Week 28; n= 10 | 3.0478 (73.2)
  CD19+CD27+IgD-; Week 104; n= 10: number analyzed (Participants) | 10
  CD19+CD27+IgD-; Week 104; n= 10 | 1.3051 (147.1)
  CD19+CD27+IgD-; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD19+CD27+IgD-; 6 month follow up; n= 7 | 0.3440 (163.8)
  CD4+ CD25hi CD45RA- IL7Rhi; Week 8; n= 12: number analyzed (Participants) | 12
  CD4+ CD25hi CD45RA- IL7Rhi; Week 8; n= 12 | 0.7010 (86.7)
  CD4+ CD25hi CD45RA- IL7Rhi; Week 16; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi CD45RA- IL7Rhi; Week 16; n= 10 | 0.5340 (221.3)
  CD4+ CD25hi CD45RA- IL7Rhi; Week 28; n= 9: number analyzed (Participants) | 9
  CD4+ CD25hi CD45RA- IL7Rhi; Week 28; n= 9 | 0.5718 (669.2)
  CD4+ CD25hi CD45RA- IL7Rhi; Week 104; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi CD45RA- IL7Rhi; Week 104; n= 10 | 4.1865 (509.4)
  CD4+ CD25hi CD45RA- IL7Rh; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD4+ CD25hi CD45RA- IL7Rh; 6 month follow up; n= 7 | 1.8067 (1456.7)
  CD4+ CD45RA- IL-7Rhi; Week 8; n= 12: number analyzed (Participants) | 12
  CD4+ CD45RA- IL-7Rhi; Week 8; n= 12 | 1.4174 (19513.4)
  CD4+ CD45RA- IL-7Rhi; Week 16; n= 10: number analyzed (Participants) | 10
  CD4+ CD45RA- IL-7Rhi; Week 16; n= 10 | 1.8613 (99527.6)
  CD4+ CD45RA- IL-7Rhi; Week 28; n=9: number analyzed (Participants) | 9
  CD4+ CD45RA- IL-7Rhi; Week 28; n=9 | 2.8378 (49940.7)
  CD4+ CD45RA- IL-7Rhi; Week 104; n= 10: number analyzed (Participants) | 10
  CD4+ CD45RA- IL-7Rhi; Week 104; n= 10 | 0.1517 (33534.3)
  CD4+ CD45RA- IL-7Rhi; 6 month follow-up; n= 7: number analyzed (Participants) | 7
  CD4+ CD45RA- IL-7Rhi; 6 month follow-up; n= 7 | 0.3532 (966.4)
  CD4+ CD25hi xIL-7Rlo; Week 8; n= 12: number analyzed (Participants) | 12
  CD4+ CD25hi xIL-7Rlo; Week 8; n= 12 | 0.7285 (85.7)
  CD4+ CD25hi xIL-7Rlo; Week 16; n= 11: number analyzed (Participants) | 11
  CD4+ CD25hi xIL-7Rlo; Week 16; n= 11 | 0.6232 (317.6)
  CD4+ CD25hi xIL-7Rlo; Week 28; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi xIL-7Rlo; Week 28; n= 10 | 0.7010 (961.5)
  CD4+ CD25hi xIL-7Rlo; Week 104; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi xIL-7Rlo; Week 104; n= 10 | 3.1025 (932.7)
  CD4+ CD25hi xIL-7Rlo; 6 month follow-up; n= 7: number analyzed (Participants) | 7
  CD4+ CD25hi xIL-7Rlo; 6 month follow-up; n= 7 | 2.0827 (832.7)
  CD4+ CD25hi IL-7Rlo; Week 8; 12: number analyzed (Participants) | 12
  CD4+ CD25hi IL-7Rlo; Week 8; 12 | 2.3001 (29702.5)
  CD4+ CD25hi IL-7Rlo; Week 16; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi IL-7Rlo; Week 16; n= 10 | 2.9023 (136702.6)
  CD4+ CD25hi IL-7Rlo; Week 28; n= 9: number analyzed (Participants) | 9
  CD4+ CD25hi IL-7Rlo; Week 28; n= 9 | 3.3453 (35372.4)
  CD4+ CD25hi IL-7Rlo; Week 104; n= 10: number analyzed (Participants) | 10
  CD4+ CD25hi IL-7Rlo; Week 104; n= 10 | 0.3410 (72506.2)
  CD4+ CD25hi IL-7Rlo; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD4+ CD25hi IL-7Rlo; 6 month follow up; n= 7 | 0.9978 (32.7)
  CD4+ CD45RA-; Week 8; n= 12: number analyzed (Participants) | 12
  CD4+ CD45RA-; Week 8; n= 12 | 0.7532 (44.5)
  CD4+ CD45RA-; Week 16; n= 11: number analyzed (Participants) | 11
  CD4+ CD45RA-; Week 16; n= 11 | 0.7638 (55.4)
  CD4+ CD45RA-; Week 28; n= 10: number analyzed (Participants) | 10
  CD4+ CD45RA-; Week 28; n= 10 | 0.9032 (71.1)
  CD4+ CD45RA-; 104; n= 10: number analyzed (Participants) | 10
  CD4+ CD45RA-; 104; n= 10 | 0.9750 (95.8)
  CD4+ CD45RA-; 6 month follow up; n= 7: number analyzed (Participants) | 7
  CD4+ CD45RA-; 6 month follow up; n= 7 | 1.0792 (90.0)

39. Secondary Outcome: Change From Baseline in Cytokines/Chemokine
Description: Cytokine/chemokine associated with T helper skewing or autoimmune pathology will be analyzed using Luminex, ELISA. Serum analyte quantification were used to confirm altered protein levels of any gene expression increases or decreases identified by transcriptomic analysis. Endpoint was moved to 'Exploratory' in Protocol amendment 5 as benefits of assessing cytokines was deemed low. Samples were not analyzed.
Time Frame: Baseline and up to Week 104/4 week post last dose
Population: ITT Population
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0

40. Secondary Outcome: Serum BLys Levels
Description: Free BLyS protein were analyzed using an ELISA. Serum samples were collected before treatment and after belimumab washout at Week 0 and Week 116/16 week follow-up visit.
Time Frame: Baseline and Week 116/16 week follow-up visit
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 14
pg/mL
  Day 0; n= 14 | 969.9595 (16.8)
  16 week follow up; n= 8: number analyzed (Participants) | 8
  16 week follow up; n= 8 | 12357.5558 (123.3)

41. Secondary Outcome: Urine BLys Levels as a Ratio to Creatinine
Description: B lymphocyte stimulator (BLyS) normalized by creatinine as a ratio of BLyS: creatinine. Free BLyS protein is being analyzed using an ELISA. Urine samples are being collected before treatment and after belimumab washout at Week 0 and Week 116/16 week follow-up visit. Only raw BLyS values available and unable to be assessed due to lack of comparison to a creatinine as a urine concentration marker.
Time Frame: Baseline and Week 116/16 week follow-up visit
Population: ITT Population
Arm/Group | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious adverse events (AEs) are presented from the start of study treatment up to end of study.
Description: On-therapy SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants who received at least one dose of investigational drug.
Arm/Group | Belimumab 10 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10 mg/kg IV (N=14)
Cellulitis (Infections and infestations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10 mg/kg IV (N=14)
Upper respiratory tract infection (Infections and infestations) | 6 (10)
Cellulitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (4)
Rhinitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (7)
Dizziness (Nervous system disorders) | 2 (3)
Migraine (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (3)
Chest pain (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Blood parathyroid hormone increased (Investigations) | 1 (1)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.